

#### STATISTICAL ANALYSIS PLAN

## STUDY TITLE:

An Open-label, Single-center, Three-part Study in Healthy Subjects to Investigate the Effect of Givinostat on the Pharmacokinetics of Midazolam and Dabigatran, the Effect of Clarithromycin on the Pharmacokinetics of Givinostat and the Pharmacokinetics of Single and Multiple Doses of Givinostat.

Protocol Code: ITF/2357/55

Type: Interventional, Pharmacokinetic and Drug-Drug Interaction

Trial

EudraCT No.: 2021-005756-11

Version: 1.0

Date of SAP: 24MAR2022

Supersedes Version: None

Date of Superseded Version: Not applicable

Sponsor: ITALFARMACO S.p.A

Via dei Lavoratori, 54

20092 Cinisello Balsamo (MI), Italy

with its registered office at Viale Fulvio Testi, 330,

Milan (MI), Italy www.italfarmaco.com Phone: + 39 02 64431 Fax: + 39 02 644346

Clinical Pharmacology Unit:

PPD

#### CONFIDENTIALITY DISCLAIMER

This document is confidential and is available for review to investigators, regulatory bodies and study audit personnel. No part of this document may be used, published, copied or otherwise disclosed without prior written authorization from PPD

or the Sponsor of this study.

1.2.



Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 1. SIGNATURE PAGE

# 1.1. Clinical Research Unit

| PPD , PharmD, MSc, PhD<br>Head of Pharmacometrics | | |
|---------------------------------------------------|-----------|------|
| PPD PPD | Signature | Date |
| PPD , MD, PhD<br>Clinical Pharmacology Director | | |
| PPD | Signature | Date |
| PPD | | |
| Sponsor's Representative | | |
| PPD , MD | | |
| Clinical R&D Director | | |
| Italfarmaco S.p.A. | Signature | Date |
| PPD | | |



# 2. CONTENTS AND ABBREVIATIONS

# 2.1. Table of Contents

| 1. | SIGNATURE PAGE | . 2 |
|---|---|---|
| | 1.1. CLINICAL RESEARCH UNIT | . 2 |
| | 1.2. Sponsor's Representative | . 2 |
| 2. | CONTENTS AND ABBREVIATIONS | . 3 |
| | 2.1. TABLE OF CONTENTS | . 3 |
| | 2.2. List of Abbreviations | . 5 |
| 3. | INTRODUCTION | . 8 |
| 4. | STUDY OBJECTIVES | . 8 |
| | 4.1. Primary | . 8 |
| | 4.2. Secondary | . 8 |
| 5. | INVESTIGATIONAL PLAN | . 8 |
| | 5.1. STUDY DESIGN | . 8 |
| | 5.1.1. Rational for Study Design | |
| | 5.1.2. Rational for Dose Selection and Treatment Duration | |
| | 5.2. STUDY PLAN | |
| | 5.2.1. Part 1 – Inhibitory and Inducing Effect of Oral Givinostat on the Single 1 | |
| | Pharmacokinetics of Intravenous and Oral Midazolam | |
| | 5.3.1. Part 1 | |
| | 5.4. RANDOMIZATION | |
| | 5.5. BLINDING | |
| | 5.6. STATISTICAL HYPOTHESIS | |
| | 5.6.1. Part 1 | 11 |
| 6. | STUDY ASSESSMENTS | 12 |
| | 6.1. SAFETY ASSESSMENTS | 12 |
| | 6.1.1. Medical History | |
| | 6.1.2. Physical Examination | |
| | 6.1.3. Weight, Height and Body Mass Index | |
| | 6.1.4. Vital Signs | |
| | 6.1.6. Laboratory Safety Tests | |
| | 6.1.7. Adverse Events | |
| | 6.1.8. Previous and Concomitant Medications | |
| | 6.2. PHARMACOKINETIC ASSESSMENTS | |
| | 6.2.1. Blood Sampling for Pharmacokinetic Assessments | |
| | 6.2.2. Plasma Pharmacokinetic Parameters | 17 |
| 7. | STUDY ENDPOINTS | 18 |
| | 7.1. Primary | 18 |
| | 7.2. Secondary | 18 |

| • | ANALYSIS POPULATIONS | 19 |
|---|---|---|
| | 8.1. PART 1 | 19 |
| | 8.1.1. Part 1 Safety Analysis Population | |
| | 8.1.2. Part 1 Pharmacokinetic Analysis Population | |
| | 8.1.3. Part 1 Drug-Drug Interaction Comparable Bioavailability Analys. | |
| | Populations | 19 |
| | DATA REVIEW / TRANSFORMATION | 20 |
| | 9.1. Data Management | 21 |
| | 9.2. ACCEPTANCE OF DATA | |
| | 9.3. Data Transformation (CDISC) | 21 |
| | STATISTICAL METHODS | 23 |
| | 10.1. GENERAL CONSIDERATIONS | 23 |
| | 10.2. Subjects' Disposition | 23 |
| | 10.3. PROTOCOL DEVIATIONS | |
| | 10.4. PLASMA PHARMACOKINETIC CONCENTRATIONS | |
| | 10.5. PLASMA PHARMACOKINETIC PARAMETERS | |
| | 10.6. Drug-Drug Interaction Comparative Bioavailability Statistic | |
| | ANALYSIS | |
| | 10.6.1. Part 1 | |
| | 10.7. SAFETY DATA ANALYSIS | |
| | PRESENTATION OF RESULTS | 26 |
| | 11.1. STATISTICAL OUTPUT SPECIFICATION | |
| | 11.2. PLANNED TABLES, FIGURES, AND SUBJECT DATA LISTINGS | |
| | 11.2.1. In-text Tables and Figures | |
| | 11.2.2. Tables, Figures and Graphs Referred to But Not Included in the | |
| | 14 of CSR) | |
| | 11.2.3. List of Subject Data Listings (Section 16.2 of CSR) | |
| | REFERENCES | 47 |
| | APPENDICES | 48 |
| | APPENDIX A. PLANNED TABLES, FIGURES, AND SUBJECT DATA LISTINGS | 48 |
| | A.1. In-text Tables and Figures – For CSR Synopsis | |
| | A.2. In-text Tables and Figures – For CSR Body Text | 61 |
| | A.3. Tables, Figures and Graphs Referred to But Not Included in the Text | (Section 14 |
| | of CSR) | |
| | A.4. List of Subject Data Listings (Section 16.2 of CSR) | 102 |
| | ANNEXES | 137 |

#### 2.2. List of Abbreviations

α Type I Error (Significance Level)

Ab Antibody

ADaM Analysis Data Model

ADAMIG Analysis Data Model Implementation Guide
ADPC Analysis Data Pharmacokinetic Concentrations
ADPP Analysis Data Pharmacokinetic Parameters

ADSL Subject-Level Analysis

AE Adverse Event
ALP Alkaline Phosphatase
ALT Alanine Aminotransferase

A<sub>mean</sub> Arithmetic Mean ANOVA Analysis of Variance

aPTT Activated Partial Thromboplastin Time

AST Aspartate Aminotransferase ATC Anatomic Therapeutic Chemical

AUC Area Under the Concentration Versus Time Curve

AUC<sub>0-t</sub> AUC from Time Zero to Last Sampling Time with Quantifiable Concentrations

 $AUC_{0-\infty}$  AUC from Time Zero to Infinity

AUC<sub>0-r,ss</sub> AUC Corresponding to the Dosing Interval, at Steady State

AURC<sub>0-t</sub> Area Under the Urinary Excretion Rate Curve from Time 0 to the Last Rate

%AUC<sub>extrap</sub> Residual Area or Percentage of Extrapolated Part of AUC<sub>0-∞</sub>

BDS Basic Data Structure

BLQ Below the Limit of Quantification

BMI Body Mass Index
bpm Beats Per Minute
Co Pre-dose Concentration
CI Confidence Interval
Cl Total Body Clearance
CK Creatine Kinase

Cl/F Total Body Clearance Affected by the Bioavailability Factor

Cl<sub>R</sub> Renal Clearance

Cl<sub>R</sub>/F Renal Clearance Affected by the Bioavailability Factor

C<sub>last</sub> Last Quantifiable Concentration C<sub>max</sub> Maximum Observed Concentration

C<sub>max.ss</sub> Maximum Observed Plasma Concentration at Steady State

Cr<sub>CL</sub> Creatinine Clearance
CSP Clinical Study Protocol
CSR Clinical Study Report
CV% Coefficient of Variation
CYP Cytochrome P450
DBP Diastolic Blood Pressure
DDI Drug-Drug Interaction

DM Demographics ECG Electrocardiogram F Bioavailability Factor

FDA Food and Drug Administration GGT Gamma-Glutamyltransferase GLP Good Laboratory Practices



Statistical Analysis Plan

Geometric Mean Gmean

Geometric Least Square Means Ratio **GMR** Geometric Coefficient of Variation GCV% GSD Geometric Standard Deviation

**Null Hypothesis**  $H_0$ Alternative Hypothesis  $H_1$ HBsAg Hepatitis B Surface Antigen Human Chorionic Gonadotropin hCG Hepatitis C Virus Antibodies **HCVAb** HIV Human Immunodeficiency Virus

ICH International Conference on Harmonization

International Normalized Ratio **INR** ISCV% Intra-Subject Coefficient of Variation

IV Intravenous

LC-MS/MS Liquid Chromatography with Tandem Mass Spectrometry

Lactate Dehydrogenase LDH Lower Limit of Quantification LLOQ

**LSmeans** Least Square Means

Mean Corpuscular Hemoglobin **MCH** 

Mean Corpuscular Hemoglobin Concentration MCHC

Mean Corpuscular Volume **MCV** 

Medical Dictionary for Regulatory Activities MedDRA

MSE Mean Square Error Molecular Weight MW

Non-Compartmental Analysis NCA PC Pharmacokinetic Concentrations PCL Protocol Clarification Letter

P-Glycoprotein P-gp

PP Pharmacokinetic Parameters PT MedDRA Preferred Term

QTcF Corrected QT Interval by Fridericia

**RBC** Red Blood Cell

Coefficient Variation of the Red Cell Distribution Width **RDW-CV** RSQ Goodness of Fit for the Terminal Elimination Phase

Rich Text File rtf

SAE Serious Adverse Event Statistical Analysis Plan SAP Serious Adverse Reaction SAR

Severe Acute Respiratory Syndrome Coronavirus 2 SARS-CoV-2

Statistical Analysis Software SAS Systolic Blood Pressure SBP SDStandard Deviation

Study Data Tabulation Model SDTM

Study Data Tabulation Model Implementation Guide SDTMIG

MedDRA System Organ Class SOC Standard Operating Procedure SOP Treatment-Emergent Adverse Events TEAE

Tables, Figures and Listings **TFLs** 

Time to Maximum Observed Concentration Tmax

Time to Maximum Observed Concentration at Steady State  $T_{max.ss}$ 



Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

TOST Two One-Sided T-Tests
TSH Thyroid-Stimulating Hormone
t<sub>0</sub> Time of Dosing (t=0h)

t<sub>½</sub> Apparent Terminal Elimination Half-Life

ULOQ Upper Limit of Quantification V<sub>D</sub> Apparent Volume of Distribution

V<sub>D</sub>/F Apparent Volume of Distribution Affected by the Bioavailability Factor (F)

WBC White Blood Cell

WHO World Health Organization

 $\lambda_z$  Apparent Terminal Elimination Rate Constant

τ Dosing Interval

#### 3. INTRODUCTION

This Statistical Analysis Plan (SAP) details the statistical methodology to be used in analysing study data and outlines the statistical programming specifications for the Tables, Figures and Listings (TFLs). This document describes the variables and populations, anticipated data transformation and manipulations and other details of the analysis not provided in the Clinical Study Protocol (CSP).

The described analyses are based on the final CSP version 1.0, dated 29NOV2021 [1] and a Protocol Clarification Letter (PCL) dated 25FEB2022. This SAP was finalized prior to data base lock and conduct of the statistical analyses. For each part of the study at the time of the Blind Review Process, a Data Blind Review Process Minute will be prepared and attached to this document (Annex 1).

Additional pharmacokinetic and statistical analysis may be performed to supplement the planned analyses described in this SAP. These supplemental analyses will be identified and presented in the Clinical Study Report (CSR).

#### 4. STUDY OBJECTIVES

## 4.1. Primary

- 1. To assess the potential inhibitory and inducing effect of oral givinostat on the single dose pharmacokinetics of intravenous (IV) and oral midazolam (Part 1).
- 2. To assess the potential inhibitory and inducing effect of oral givinostat on the single dose pharmacokinetics of oral dabigatran etexilate (Part 1).

## 4.2. Secondary

1. To assess the safety and tolerability of concomitant administration of givinostat plus midazolam and dabigatran etexilate (Part 1).

## 5. INVESTIGATIONAL PLAN

# 5.1. Study Design

This is a phase I, open-label, 3-part, fixed-sequence, non-randomized study in healthy male and female subjects.

Study parts may be conducted concomitantly.

# 5.1.1. Rational for Study Design

The rational for study design detailed in the CSP [1].

In Part 1, the perpetrator drug-drug interaction (DDI) potential of givinostat as inhibitor and inducer of cytochrome P450 (CYP)3A and P-glycoprotein (P-gp) activity will be evaluated.

## 5.1.2. Rational for Dose Selection and Treatment Duration

#### 5.1.2.1. Part 1

## Rationale for Givinostat Dose and Treatment Duration as Perpetrator

A dose of 50 mg givinostat will be administered twice-daily to subjects in order to maximize the possibility to identify a DDI with midazolam and dabigatran etexilate. The inhibitory effect will be assessed on Days 6 to 9 and the inducing effect will assessed on Days 17 to 20 [1].

## Rationale for Substrates Dose

To access a DDI at CYP3A4 level, a therapeutic single-dose of 1 mg midazolam IV, and 2.5 mg single-dose of oral midazolam will be administered, in the present study.

To access a DDI at P-gp level, a therapeutic single-dose of 75 mg dabigatran will be administered [1].

# Rationale for Perpetrator and Substrates Administration Schedule

In order to potentiate the maximal P-gp and CYP3A inhibition by the perpetrator, midazolam and dabigatran administration will occur 1 hour after the givinostat morning dose on Days 6, 7, 17 and 18 [1].

#### 5.2. Study Plan

# 5.2.1. Part 1 – Inhibitory and Inducing Effect of Oral Givinostat on the Single Dose Pharmacokinetics of Intravenous and Oral Midazolam

Subjects will be confined in BlueClinical Phase I from Day -1 to Day 20.

On Days 1, 6 and 17, single doses of midazolam 1 mg IV and dabigatran etexilate 75 mg, will be administered 1 hour after the planned morning time of givinostat administration.

On Days 2, 7 and 18, a single oral dose of midazolam 2.5 mg oral solution will be administered 1 hour after the planned morning time of givinostat administration.

From Day 4 to Day 18, givinostat 50 mg as oral suspension will be administered twice a day, in the morning and in the evening. On Day 19, only the morning dose will be administered.

Midazolam and dabigatran etexilate will be administered following an overnight fasting of at least 8 hours and subjects will remain fasted until at least 3 hours post-dose. Oral midazolam and dabigatran etexilate will be administered with 150 mL of water. Except for water given with the investigational products, no fluids will be allowed from 1 hour before midazolam and dabigatran dosing until 2 hours post dose. Water will be provided ad libitum at all other times.

Midazolam and dabigatran etexilate will be administered with the subjects in a semi-recumbent position. Subjects will remain semi-recumbent until at least 3 hours post-dose.

The following assessments will be performed:

- Blood collection for pharmacokinetic analysis on Days 1 to 4, 6 to 9 and 17 to 20.
- Vital signs measurements (blood pressure [BP], pulse rate [PR] and respiratory rate [RR]) on Days 1, 2, and 4 to 19.

- 12-lead electrocardiogram (ECG) on Days 3 to 19.
- Blood collection for laboratory tests (hematology, biochemistry and coagulation on Days 4 and 9 and hematology on Days 6, 12, 15 and 18).

Subjects will be discharged from BlueClinical Phase I in the morning of Day 20 if allowed by the investigator based on their medical condition. The following procedures will be performed:

- Physical examination.
- Collection of body weight.
- Vital signs measurements (BP, PR, RR and body temperature).
- 12-lead ECG.
- Safety laboratory assessments (hematology, biochemistry, coagulation and urinalysis).
- Serum pregnancy test for all female subjects.

Subjects will return to BlueClinical Phase I 10 to 14 days after the end of study to undergo additional assessments as required per protocol.

The total duration of Part 1 for each subject will be up to approximately 8 weeks from Screening to Follow-up visit, divided as follows:

- Screening: up to 21 days
- Treatment Period: Days 1 to 20
- Safety follow-up visit: 12±2 days

## 5.3. Number of Participants and Sample Size Estimation

To ensure enough subjects with evaluable data complete each study part, a total of fifty-four (54) healthy male and female subjects are planned to be enrolled as follows:

- Part 1: twenty-six (26) subjects
- Part 2: twenty (20) subjects
- Part 3: eight (8) subjects

Each subject will participate in one study part only.

#### 5.3.1. **Part 1**

<u>Midazolam</u>: Assuming an Intra-Subject Coefficient of Variation (ISCV%) of  $\leq$ 23% for midazolam  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$ , a true geometric means ratio (midazolam with vs without givinostat) of 1.00, a significance level (alpha error) of 5%, and a default no-effect boundary of 80.00% to 125.00%, a sample of 20 evaluable subjects results in at least 80% power. Accounting for early-termination subjects, a sample size of 26 subjects will be enrolled.

<u>Dabigatran</u>: Assuming an ISCV% of approximately 30% for dabigatran  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$ , a true geometric means ratio (dabigatran with vs without givinostat) of 1.00, a significance level (alpha error) of 5%, and that the two-sided 90% confidence interval (CI) for the geometric means ratio of  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-\infty}$  will lie within 74.62% to 134.02%, a sample of 20 evaluable subjects results in at least 80% power. Accounting for early-termination subjects, a sample size of 26 subjects will be enrolled.

## 5.4. Randomization

This is a fixed sequence study. Randomization is not applicable.

# 5.5. Blinding

The study will be conducted as open label. Blinding procedures are not applicable.

# 5.6. Statistical Hypothesis

#### 5.6.1. Part 1

Part 1 of the study is designed to:

- 1. assess the potential inhibitory and inducing effect of oral givinostat on the single dose pharmacokinetics of IV and oral midazolam.
- assess the potential inhibitory and inducing effect of oral givinostat on the single dose pharmacokinetics of oral dabigatran etexilate.

As in accordance with FDA Guidance on DDI studies [2], assessment of DDI will be based upon the 90% confidence interval (CI) for the Geometric Least Square Means (LSmeans) Ratio (GMR) for the primary pharmacokinetic parameters.

This method is equivalent to two one-sided t-tests (TOST) with the null hypothesis ( $H_0$ ) of non-comparable bioavailability at the 5% significance level ( $\alpha = 0.05$ ).

For midazolam, assuming a maximum 20% difference between midazolam co-administered with givinostat and administered alone, the interval hypotheses for comparable bioavailability can be formulated as:

$$H_0:~\mu_T/\mu_R < 0.80~~\text{or}~~\mu_T/\mu_R > 1.25$$
 versus  $~H_1:~~0.80 \le \mu_T/\mu_R \le 1.25$ 

where  $\mu_T$  and  $\mu_R$  are the Geometric LSmeans for midazolam co-administered with givinostat and administered alone, respectively.

Hence, the hypothesis is to show comparable bioavailability by rejecting the  $H_0$  of non-comparable bioavailability, i.e., the decision of comparable bioavailability is made based on whether the 90% CI of the midazolam co-administered with givinostat-to-midazolam administered alone GMR is within 80.00 - 125.00% [2].

For dabigatran, assuming a maximum 25.38% difference between midazolam co-administered with givinostat and administered alone, the interval hypotheses for comparable bioavailability can be formulated as:

where  $\mu_T$  and  $\mu_R$  are the Geometric LSmeans for dabigatran co-administered with givinostat and administered alone, respectively.

Hence, the hypothesis is to show comparable bioavailability by rejecting the  $H_0$  of non-comparable bioavailability, i.e., the decision of comparable bioavailability is made based on whether the 90% CI of the dabigatran co-administered with givinostat-to-dabigatran administered alone GMR is within 74.62 - 134.02% [2].

#### 6. STUDY ASSESSMENTS

For each study part, a summary of procedures for study assessments are presented in Section 2 of the CSP (Study Flow-Chart and Study Design Diagram) [1].

# 6.1. Safety Assessments

Subjects' safety will be monitored during the study.

Safety assessments will include pre-study medical history, physical examination, vital signs, 12-lead ECG, clinical laboratory tests and adverse event (AE) monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety.

Medications will be mentioned according to the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system.

# 6.1.1. **Medical History**

Medical history will cover all relevant past or present information related to subject's health at the time of informed consent signature.

Medical history at screening will include past or present relevant cardiovascular, respiratory, renal, genitourinary, gastrointestinal, hepatic, hematological, immunological, endocrine, dermatological, musculoskeletal, neurological, psychiatric, drug and surgical history, or any other diseases or disorders.

Medical history will be referred in accordance with the Medical Dictionary for Regulatory Activities (MedDRA), version 24.1 or higher.

Adverse events related to medical history will be identified.

#### 6.1.2. Physical Examination

Physical examination at screening and end-of-study will include: general appearance; skin; head and neck; thorax and abdomen; pulmonary auscultation; cardiac auscultation; abdomen palpation; limbs; brief neurological examination.

# 6.1.3. Weight, Height and Body Mass Index

The body height and weight values as well as the body mass index (BMI) will be recorded in the electronic case report form (eCRF) and will be determined at Screening. Only body weight will be

determined also at admission and end-of-study.

The subjects' body weight will preferably be measured using the same weighing scale for all subjects and throughout the study. The weighing scale should have a precision of at least 0.5 kg.

## 6.1.4. Vital Signs

Vital signs will include:

- Systolic blood pressure (SBP).
- Diastolic blood pressure (DBP).
- Pulse rate (PR).
- Respiratory rate (RR).
- Body temperature.

# 6.1.5. 12 Lead Electrocardiogram

A 12-lead ECG will be performed preferably before the blood collection. The corrected QT interval by Fridericia (QTcF) will be analyzed.

# 6.1.6. Laboratory Safety Tests

The following laboratory parameters will be tested:

- Hematology:
  - Red blood cell (RBC) count.
  - White blood cell (WBC) count.
  - WBC differential count:
    - Neutrophils.
    - Eosinophils.
    - Basophils.
    - Lymphocytes.
    - Monocytes.
  - Hemoglobin.
  - Mean corpuscular volume (MCV).
  - Mean corpuscular hemoglobin (MCH).
  - Mean corpuscular hemoglobin concentration (MCHC).
  - Coefficient variation of the red cell distribution width (RDW-CV).
  - Hematocrit.
  - Platelet count.
  - Mean platelet volume.
- Coagulation:
  - Prothrombin rate.
  - Prothrombin time.
  - Prothrombin time international normalized ratio (INR).
  - Activated partial thromboplastin time (aPTT).
- General biochemistry:
  - Total bilirubin.
  - Direct bilirubin.
  - Indirect bilirubin.

- Alkaline phosphatase (ALP).
- Amylase.
- Aspartate aminotransferase (AST).
- Alanine aminotransferase (ALT).
- Lactate dehydrogenase (LDH).
- Cystatin C.
- C-reactive protein.
- Gamma-glutamyltransferase (GGT).
- Creatinine kinase (CK).
- Total protein.
- Albumin.
- Uric acid.
- Triglycerides.
- Total cholesterol.
- Low-density lipoprotein-cholesterol (LDL-C).
- High-density lipoprotein-cholesterol (HDL-C).
- Sodium.
- Potassium.
- Chloride.
- Calcium.
- Magnesium.
- Glucose.
- Creatinine.
- Urea.
- Thyroid-stimulating hormone (TSH).
- Estimated creatinine clearance (Cr<sub>CL</sub>).
- Viral Serology:
  - Human Immunodeficiency Virus (HIV):
    - HIV-1 (anti-HIV-1Ab).
    - HIV-2 (anti-HIV-2Ab).
  - Hepatitis B (HBsAg)
  - Hepatitis C (anti-HCVAb).
- Beta-human chorionic gonadotropin (beta-hCG) pregnancy tests:
  - Serum.
  - Urine.
- Urinalysis:
  - · рН.
  - Specific gravity.
  - Protein.
  - Hemoglobin.
  - Glucose.
  - Ketones.
  - Bilirubin.
  - Nitrites.
  - Urobilinogen.
  - Microscopy.
- Drugs-of-abuse urine test:

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- Cannabinoids.
- Opiates.
- Cocaine.
- Amphetamines.
- Benzodiazepines.
- Ethanol urine test.
- Cotinine urine test.
- Follicle-stimulating hormone (FSH) test.
- Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) diagnostic tests.

#### 6.1.7. Adverse Events

The occurrence of clinical AEs will be monitored throughout the study.

Clinically significant abnormalities in laboratory safety tests, vital signs and physical examination will be reported as AEs.

Treatment-emergent AEs (TEAEs) are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the subject receives the first dose of investigational product. TEAEs that occur after administration of investigational product during the washout of a given period will be assigned to the treatment administered in that period.

The following information will be used for the description of the AEs:

- Reported Term.
- Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) coding.
- MedDRA Preferred Term (PT) coding.
- Start date and time.
- End date and time.
- Seriousness.
- Severity:
  - Mild.
  - Moderate.
  - Severe.
- Relationship (causality) for each treatment administrated, per part.
  - Reasonably Possible.
  - Not Reasonably Possible.
  - Unknown.
- Action taken:
  - Dose Increased.
  - Dose Not Changed.
  - Dose Rate Reduced.
  - Dose Reduced.
  - Drug Interrupted.
  - Drug Withdrawn.
  - Not Applicable.
  - Unknown.

- Concomitant medication.
- Outcome:
  - Fatal.
  - Not Recovered / Not Resolved.
  - Recovered / Resolved.
  - Recovered / Resolved with Sequelae.
  - Recovering / Resolving.
  - Unknown.
- Most recent study treatment taken.
- Last dosing date.

#### 6.1.8. Previous and Concomitant Medications

A previous medication is any medication for which the end date is prior to first dosing. A concomitant medication is any medication ongoing or initiated after first dosing.

For all study parts, the use of any medications including Over-the-Counter (OTC) products (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) is forbidden from 28 days or within 5 half-lives of the medicinal product, whichever is longer, prior to admission up to last sample for pharmacokinetics assessment, except for medications for the treatment of AEs.

In study Part 1, the use of anticoagulants is forbidden within 28 days or 5 drug half-lives, whichever is longer, prior to admission until the end of study.

Any medication (previous or concomitant) taken within the period of medication restriction must be recorded in the eCRF. If concomitant medication is ongoing at the follow-up visit, no end date will be provided in the eCRF.

For each study part, previous and concomitant medications used by study participants during the study and their judged impact on the pharmacokinetic assessment will be listed in the respective Data Blind Review Meeting/ Process Minute (Annex 1).

Concomitant medications will be coded according to the WHO ATC classification system.

#### 6.2. Pharmacokinetic Assessments

# 6.2.1. Blood Sampling for Pharmacokinetic Assessments

In each study part, while subject is confined at the clinical research unit, blood samples will be taken preferably via an indwelling cannula placed in a vein of an upper limb of the subject. During ambulatory visits, blood samples will be taken by direct venipuncture.

The actual time of all pharmacokinetic blood draws will be recorded and reported for all subjects. The pre-dose blood sample will be collected within 30 minutes before dosing. The post-dose blood samples will be collected within  $\pm 3$  minutes from the scheduled sampling time. Greater deviations will be reported as a protocol deviation and its cause will be recorded.



In case blood sampling for pharmacokinetics and other procedures coincide in time, blood draws will have priority unless other procedures are necessary for assuring subject's safety.

will carry out the determination of plasma levels of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563), midazolam, 1-hydroxymidazolam and total and free dabigatran in accordance with the applicable principles of Good Laboratory Practices (GLP), using a previously validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) analytical method.

The planned lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for:

- givinostat are 1 and 100 ng/mL.
- givinostat metabolite ITF2374 are 1 and 100 ng/mL.
- givinostat metabolite ITF2375 are 1 and 100 ng/mL.
- givinostat metabolite ITF2440 are 10 and 500 ng/mL.
- givinostat metabolite ITF2563 are 2 and 125 ng/mL.
- midazolam are 100 and 100000 pg/mL.
- 1-hydroxymidazolam are 100 and 50000 pg/mL.
- total dabigatran are 1 and 400 ng/mL.
- free dabigatran are 1 and 400 ng/mL.

LLOQ represents a value lower than or equal to 1/20 of estimated  $C_{\text{max}}$  value. Any adjustment to this range will be documented in the study specific Bioanalytical Report, which will supersede the indicated range.

#### 6.2.1.1. Part 1

A total of one hundred and seventeen (117) blood samples will be collected as follows:

- Thirteen (13) blood samples of 3 mL each will be collected in K<sub>2</sub>-EDTA collection tubes at pre-dose and at 2 minutes, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12 and 24 hours after the administration of midazolam IV, on Days 1, 6 and 17, for the determination of midazolam and 1-hydroxymidazolam plasma concentrations.
- Eleven (11) blood samples of 3 mL each will be collected in K<sub>2</sub>-EDTA collection tubes at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hours after the administration of oral midazolam, on Days 2, 7 and 18, for the determination of midazolam and 1-hydroxymidazolam plasma concentrations. The 24-hour blood collection following midazolam IV will be assumed as the pre-dose sampling for oral midazolam.
- Fifteen (15) blood samples of 4 mL each will be collected in K<sub>2</sub>-EDTA collection tubes at pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after the administration of dabigatran etexilate, on Days 1, 6 and 17, for the determination of total and free dabigatran plasma concentrations.

#### 6.2.2. Plasma Pharmacokinetic Parameters

The following pharmacokinetic parameters will be derived by standard non-compartmental analysis (NCA) methods from the single-dose plasma concentration *versus* time profiles, for:

- Part 1:
  - midazolam.
  - 1-hydroxymidazolam.
  - total dabigatran.

# free dabigatran.

| Parameter | Description |
|---|---|
| $C_{max}$ | Maximum observed concentration, directly obtained from the observed concentration <i>versus</i> time profile. |
| $T_{\text{max}}$ | Time of occurrence of maximum observed concentration. |
| AUC <sub>0-t</sub> <sup>1</sup> | Area under the concentration <i>versus</i> time curve (AUC) from time of dosing (t=0h) to the time of the last measurable concentration (t <sub>last</sub> ), calculated by the linear-up/log-down trapezoidal method. |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Total AUC extrapolated to infinity, calculated as $AUC_{0-t} + \frac{C_{last}}{\lambda_{\sigma}}$ , where $C_{last}$ |
| | is the last measurable concentration and $\lambda_z$ is the apparent terminal elimination rate constant. |
| %AUC <sub>extrap</sub> | Percentage of $AUC_{0-\infty}$ due to extrapolation from the time of the last measurable concentration (t <sub>last</sub> ) to infinity, i.e., residual area, calculated as $100 \cdot \frac{AUC_{0-\infty} - AUC_{0-t}}{AUC_{0-\infty}}$ . |
| $\lambda_{\mathbf{z}}$ | Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration <i>versus</i> time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations. |
| t <sub>1/2</sub> | Apparent terminal elimination half-life, calculated as $\frac{ln(2)}{\lambda_{-}}$ . |

 $<sup>^{1}</sup>$  In Part 1, for midazolam and its metabolite the last sampling time corresponds to 24 hours, and for total and free dabigatran the last sampling time corresponds to 72 hours.

The upper and the lower timepoints and the number of timepoints used for  $\lambda_z$  estimation, as well as the goodness of fit for the terminal elimination phase (RSQ), will be reported. No values of  $\lambda_z$ , AUC<sub>0-∞</sub>, %AUC<sub>extrap</sub> and t<sub>½</sub> will be reported for cases where  $\lambda_z$  cannot be reliably determined.

## 7. STUDY ENDPOINTS

# 7.1. Primary

1. Midazolam and dabigatran plasma concentrations and thereof derived pharmacokinetic parameters alone and in combination with givinostat (Part 1).

# 7.2. Secondary

 Incidence and severity of AEs; changes in vital signs, physical examination, ECG and clinical laboratory tests following administration of midazolam and dabigatran etexilate alone and in combination with givinostat (Part 1).

#### 8. ANALYSIS POPULATIONS

The analysis populations are defined in accordance with the CSP [1].

For each study part, the subjects to be included in each analysis population will be reported in the respective Data Blind Review Process Minute (Annex 1).

For each study part, explanation of the reasons for exclusion of subjects from any analysis population will be provided in the respective Data Blind Review Process Minute (Annex 1) and in the CSR.

The list of subjects who complete each study part will be presented in Annex 2,.

#### Part 1

#### 8.1.

## Part 1 Safety Analysis Population

8.1.1.

All subjects who receive at least one dose of an IMP in Part 1 of the study will constitute the Part 1 Safety Analysis Population.

Part 1 safety data analysis will be performed for all subjects in the Part 1 Safety Analysis Population.

# Part 1 Pharmacokinetic Analysis Population

8.1.2. Part 1 Pharmacokinetic Analysis Population will include all subjects enrolled in Part 1 of the study, who are expected to provide evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation.

The following reasons justify the exclusion of the pharmacokinetic data of a subject from the Part 1 pharmacokinetic analysis population:

 Protocol violation considered to have a potentially relevant effect on the pharmacokinetic results of the study.

NOTE: These protocol violations will be reported in the Data Blind Review Process Minute (Annex 1), and their impact will be assessed at the time of pharmacokinetic analysis.

Subject experienced vomiting or diarrhea.

NOTE: Subjects that experienced vomiting or diarrhoea during this study part will be reported in the Data Blind Review Process Minute (Annex 1), and their exclusion will be assessed at the time of pharmacokinetic analysis.

- Subject with pre-dose concentration > 5% of the  $C_{\text{max}}$  value of the corresponding pharmacokinetic profile.
  - *NOTE: This exclusion will be assessed at the time of pharmacokinetic analysis.*
- Subject with lack of any measurable concentrations or only very low plasma concentrations.

NOTE: This exclusion will be assessed at the time of pharmacokinetic analysis.

#### 8.1.3. Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Populations

For each comparation of interest to assess a potential drug-drug interaction, a Drug-Drug Interaction Comparable Bioavailability Analysis Population will be defined.

# 8.1.3.1. Part 1 Inhibitory Effect of Givinostat on Midazolam IV Analysis Population

Potential Inhibitory Effect of Givinostat on Midazolam IV Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for midazolam IV administered alone (Day 1) and co-administered with givinostat (Day 6), without deviations affecting pharmacokinetic interpretation.

# 8.1.3.2. Part 1 Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population

Potential Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for oral midazolam administered alone (Day 2) and co-administered with givinostat (Day 7), without deviations affecting pharmacokinetic interpretation.

# 8.1.3.3. Part 1 Inhibitory Effect of Givinostat on Dabigatran Analysis Population

Potential Inhibitory Effect of Givinostat on Dabigatran Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for dabigatran administered alone (Day 1) and co-administered with givinostat (Day 6), without deviations affecting pharmacokinetic interpretation.

## 8.1.3.4. Part 1 Inducing Effect of Givinostat on Midazolam IV Analysis Population

Inducing Effect of Givinostat on Midazolam IV Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for midazolam IV administered alone (Day 1) and co-administered with givinostat (Day 17), without deviations affecting pharmacokinetic interpretation.

# 8.1.3.5. Part 1 Inducing Effect of Givinostat on Oral Midazolam Analysis Population

Inducing Effect of Givinostat on Oral Midazolam Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for oral midazolam administered alone (Day 2) and co-administered with givinostat (Day 18), without deviations affecting pharmacokinetic interpretation.

#### 8.1.3.6. Part 1 Inducing Effect of Givinostat on Dabigatran Analysis Population

Inducing Effect of Givinostat on Dabigatran Analysis Population will include all subjects from the Part 1 Pharmacokinetic Analysis Population who are expected to provide evaluable pharmacokinetic data for dabigatran administered alone (Day 1) and co-administered with givinostat (Day 17), without deviations affecting pharmacokinetic interpretation.

## 9. DATA REVIEW / TRANSFORMATION

# 9.1. Data Management

Data handling will be conducted in accordance with the Clinical Data Management section of the CSP and the Data Management Plan developed specifically for this study.

# 9.2. Acceptance of Data

For each study part, TFLs may start being programmed prior to or during the course of the trial. However, the programming of analysis datasets and TFLs will only be concluded and quality-controlled after database soft lock. Only audited data released by the bioanalytical laboratory will be used for programming the final analysis datasets and TFLs.

# 9.3. Data Transformation (CDISC)

Before performing the statistical analysis, all data collected (multiple sources) will be integrated into a common repository, using SAS® version 9.4 or higher.

For standardization and submission purpose, all data will be transformed according to Clinical Data Interchange Standards Consortium (CDISC):

- Study Data Tabulation Model (SDTM) version 1.4 or higher.
- SDTM Implementation Guide (SDTMIG) version 3.2 or higher.
- The following analysis datasets will be generated (Analysis Data Model [ADaM] version 2.1 or higher; ADaM Implementation Guide [ADaMIG], version 1.2 or higher) to support the results and ease the programming activities during the statistical analysis:
  - Subject-Level Analysis Dataset (ADSL).
  - Analysis Data Pharmacokinetic Concentrations (ADPC).
  - Analysis Data Pharmacokinetic Parameters (ADPP).
  - Analysis Data Adverse Events (ADAE).
  - Analysis Data Vital Signs (ADVS).
  - Analysis Data Electrocardiogram Parameters (ADEG).
  - Analysis Data Laboratory Test Results (ADLB).

For the scope of this trial, considering the primary and secondary objectives, six (6) Basic Data Structure (BDS) domains will be generated: ADPC, ADPP, ADAE, ADVS, ADEG and ADLB. These six datasets plus ADSL will be updated for each part. These domains will support the descriptive statistical analyses of the pharmacokinetic concentrations, the pharmacokinetic parameters and safety.

# ADSL - Subject-Level Analysis Dataset

This analysis domain will contain: general data about the subjects (i.e., age, sex and race), planned and actual allocated treatment analysis, and start and end dates of treatment analysis period. The origin of these data will primarily be the Demographics (DM) and Exposure (EX) SDTM domains. Besides this information, the following variables will be derived:

- Safety Population Flag Subjects included in the Safety Analysis Population.
- Pharmacokinetic Analysis Set Population Flag 1 Subjects included in the Part 1 Pharmacokinetic Analysis Population.
- Drug-Drug Interaction Analysis Set Population Flag 1 Subjects included in the Part 1
   Inhibitory Effect of Givinostat on Midazolam IV Analysis Population.



- Drug-Drug Interaction Analysis Set Population Flag 2 Subjects included in the Part 1 Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population.
- Drug-Drug Interaction Analysis Set Population Flag 3 Subjects included in the Part 1 Inhibitory Effect of Givinostat on Dabigatran Analysis Population.
- Drug-Drug Interaction Analysis Set Population Flag 4 Subjects included in the Part 1
  Inducing Effect of Givinostat on Midazolam IV Analysis Population.
- Drug-Drug Interaction Analysis Set Population Flag 5 Subjects included in the Part 1
  Inducing Effect of Givinostat on Oral Midazolam Analysis Population.
- Drug-Drug Interaction Analysis Set Population Flag 6 Subjects included in the Part 1 Inducing Effect of Givinostat on Dabigatran Analysis Population.
- Completers Population Flag Subjects who completed the treatment period.

#### ADPC – Analysis Data Pharmacokinetic Concentrations

This is a BDS dataset that will contain the concentrations for each subject, per treatment analysis, per analyte/metabolite, and per timepoint.

The origin of these data will primarily be the EX and Pharmacokinetic Concentrations (PC) SDTM domains and ADSL ADaM domain.

Besides this information, the following variables will be derived:

- Pharmacokinetic Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 1
- Drug-Drug Interaction Analysis Set Population Flag 2
- Drug-Drug Interaction Analysis Set Population Flag 3.
- Drug-Drug Interaction Analysis Set Population Flag 4.
- Drug-Drug Interaction Analysis Set Population Flag 5.
- Drug-Drug Interaction Analysis Set Population Flag 6.
- Pharmacokinetic Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 7.
- Pharmacokinetic Analysis Set Population Flag 3.
- Pharmacokinetic Analysis Set Population Flag 4.

#### ADPP – Analysis Data Pharmacokinetic Parameters

This is a BDS dataset that will contain the NCA pharmacokinetic parameters (plasma and urine) for each subject, per treatment analysis and per analyte/metabolite.

Besides the original pharmacokinetic parameter value, the dataset will contain the ln-transformed value that is necessary to apply for the specified statistical model(s).

The origin of these data will primarily be the DM and Pharmacokinetic Parameters (PP) SDTM domains.

Besides this information, the following variables will be derived:

- Pharmacokinetic Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 3.
- Drug-Drug Interaction Analysis Set Population Flag 4.
- Drug-Drug Interaction Analysis Set Population Flag 5.
- Drug-Drug Interaction Analysis Set Population Flag 6.
- Pharmacokinetic Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 7.
- Pharmacokinetic Analysis Set Population Flag 3.
- Pharmacokinetic Analysis Set Population Flag 4.



# ADAE - Analysis Data Adverse Events Dataset

This is an OCCDS dataset that will contain the adverse events for each subject.

The origin of these data will primarily be the Adverse Events (AE) SDTM domain and ADSL ADaM domain.

## ADVS – Analysis Data Vital Signs Dataset

This is a BDS dataset that will contain the vital signs results for each subject, per treatment analysis and per timepoint.

The origin of these data will primarily be the Vital Signs (VS) SDTM domain and ADSL ADaM domain.

# ADEG – Analysis Data Electrocardiogram Parameters Dataset

This is a BDS dataset that will contain the electrocardiogram for each subject, per treatment analysis and per timepoint.

The origin of these data will primarily be the ECG Test Results (EG) SDTM domain and ADSL ADaM domain.

# ADLB - Analysis Data Laboratory Test Results Dataset

This is a BDS dataset that will contain the safety laboratory test results for each subject and per treatment analysis.

The origin of these data will primarily be the Laboratory Test Results (LB) SDTM domain and ADSL ADaM domain.

## 10. STATISTICAL METHODS

#### 10.1. General Considerations

Estimation of the pharmacokinetic parameters and drug-drug interaction comparative bioavailability analysis will be conducted on Phoenix<sup>®</sup> WinNonlin<sup>®</sup> version 8.2 or higher (Certara USA Inc, Princeton, NJ). All other statistical analysis will be conducted on SAS<sup>®</sup> version 9.4 or higher.

Statistical analyses and pharmacokinetic analyses will be performed in accordance with the U.S. FDA guidances [2, 3] and BlueClinical applicable Standard Operating Procedures (SOPs).

Unless specified otherwise, continuous variables will be summarized with the following descriptive statistics: number of observations (n), mean, standard deviation (SD), minimum, median and maximum values. Categorical data will be summarized with frequencies and percentages. For subjects' characteristics and safety analyses, missing data will not be replaced; descriptive statistics and statistical analysis will be performed based on the available data only. All data recorded on discontinued subjects will be listed.

## 10.2. Subjects' Disposition

The number of subjects who completed each study part as well as subjects who withdrew prematurely from the study will be summarized by completion status and reason for withdrawal.

Subjects who prematurely withdrew from the study will be listed.

The number of subjects included in each analysis population will be summarized, for each study part.

#### 10.3. Protocol Deviations

During the respective Data Blind Review Process, all protocol deviations that occurred during each study part will be assessed in terms of their potential impact on the pharmacokinetic analysis. The result of this assessment will be reported in the respective Data Blind Review Process Minute (Annex 1).

#### 10.4. Plasma Pharmacokinetic Concentrations

For each study part (Part 1, Part 2 and Part 3), for the subjects included in the respective pharmacokinetic analysis population, descriptive statistics [n, geometric mean ( $G_{mean}$ ), arithmetic mean ( $A_{mean}$ ), SD, geometric SD (GSD), coefficient of variation (CV%), geometric CV% (GCV%), two-sided 95% CI of the  $A_{mean}$  and  $G_{mean}$ , median, minimum and maximum] of the plasma concentrations will be presented for each time point, by analyte, and by administration day. Concentrations below the LLOQ will be taken as missing for the calculation of the log-transformed statistics and as zero for the calculation of the remaining summary statistics.

For each study part (Part 1, Part 2 and Part 3), individual (per subject) and G<sub>mean</sub> (including 95% CIs) plasma concentration *versus* time profile will be graphically displayed in both linear and semi-logarithmic scales:

- For plotting individual data in linear scale, concentrations below the LLOQ will be substituted by zero.
- For plotting G<sub>mean</sub> data in linear scale, concentrations below the LLOQ will be substituted by missing.
- For plotting data in semi-logarithmic scale, concentrations below the LLOQ before t<sub>max</sub>, will be substituted by ½ of the LLOQ value. After t<sub>max</sub>, concentrations below the LLOQ will be considered as missing. However, in case of two or more consecutive concentrations below the LLOQ, the first value will be replaced by ½ of the LLOQ value and the next values will be considered as missing.

Graphic presentation of individual data will be based on actual blood sampling time, except for predose sampling time which will be assumed as t<sub>0</sub>.

Concentration data from non-evaluable periods will be listed and graphically represented separately.

#### 10.5. Plasma Pharmacokinetic Parameters

For each study part, plasma pharmacokinetic parameters will be calculated for the respective pharmacokinetic analysis population.

For each study part, for the subjects included in the pharmacokinetic analysis population, individual plasma pharmacokinetic parameters and descriptive statistics (n,  $G_{mean}$ ,  $A_{mean}$ , SD, GSD, CV%, GCV%, two-sided 95% CI of the  $A_{mean}$  and  $G_{mean}$ , median, minimum and maximum), will be presented by investigational product.

If a given pharmacokinetic parameter could not be reliably determined for more than ½ of the subjects, only the minimum and maximum values will be presented, and the other descriptive statistics will be omitted for that parameter.

Missing pharmacokinetic parameter data will not be imputed.

# 10.6. Drug-Drug Interaction Comparative Bioavailability Statistical Analysis

## 10.6.1. Part 1

Formal statistical analysis of pharmacokinetic data will be performed to characterize the following pharmacokinetic interactions:

- 1. Analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV:
  - C<sub>max</sub> and AUC<sub>0-t</sub> of midazolam and 1-hydroxymidazolam when midazolam IV is administered alone (Day 1) and co-administered with givinostat (Day 6) will be the primary pharmacokinetic parameters for the assessment of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV.
- 2. Analysis of the potential inducing effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV:
  - $C_{max}$  and  $AUC_{0-t}$  of midazolam and 1-hydroxymidazolam when midazolam IV is administered alone (Day 1) and co-administered with givinostat (Day 17) will be the primary pharmacokinetic parameters for the assessment of the potential inducing effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV.
- 3. Analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam:
  - $C_{max}$  and  $AUC_{0+}$  of midazolam and 1-hydroxymidazolam when oral midazolam is administered alone (Day 2) and co-administered with givinostat (Day 7) will be the primary pharmacokinetic parameters for the assessment of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam.
- Analysis of the potential inducing effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam:
  - C<sub>max</sub> and AUC<sub>0-t</sub> of midazolam and 1-hydroxymidazolam when oral midazolam is administered alone (Day 2) and co-administered with givinostat (Day 18) will be the primary pharmacokinetic parameters for the assessment of the potential inducing effect oral givinostat on the single-dose pharmacokinetics of oral midazolam.
- 5. Analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral dabigatran:
  - $C_{max}$  and  $AUC_{0-t}$  of total and free dabigatran when dabigatran etexilate is administered alone (Day 1) and co-administered with givinostat (Day 6) will be the primary pharmacokinetic parameters for the assessment of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral dabigatran pharmacokinetic.
- 6. Analysis of the potential inducing effect of oral givinostat on the single-dose pharmacokinetics of oral dabigatran:
  - C<sub>max</sub> and AUC<sub>0-t</sub> of total and free dabigatran when dabigatran etexilate is administered alone (Day 1) and co-administered with givinostat (Day 17) will be the primary pharmacokinetic

parameters for the assessment of the potential inducing effect of oral givinostat on the single-dose pharmacokinetics of oral dabigatran.

For each of the above comparation of interest, an analysis of variance (ANOVA) will be performed on the ln-transformed primary pharmacokinetic parameters. A linear mixed effects model will be applied, using Treatment as fixed effect, assessed at a two one-sided 5% significance level ( $\alpha = 0.05$ ). Subject will be included as random effect. Geometric least square means ratios (GMR) of the Test-to-Reference and corresponding 90% CI will be calculated for the ln-transformed primary pharmacokinetic parameters, using substrates (midazolam IV, oral midazolam, and dabigatran etexilate) co-administered with givinostat as the Test and administered alone as the Reference.

Wilcoxon signed rank test will be used to test for the difference in  $T_{max}$ . The 90% CI for median  $T_{max}$  difference will be calculated by an exact asymmetric method.

## 10.7. Safety Data Analysis

Safety and tolerability data will be listed by study part, treatment, study timepoint and subject number and summarized descriptively by study part, treatment and study timepoint.

At each time point, absolute values of safety variables and change from baseline will be summarized with mean, median, SD, SE, minimum, and maximum values. The number of available observations and absolute out-of-range values will be presented. Values outside the investigator's normal range will be flagged in the listing.

For clinical laboratory data and vital signs data, out of range values will be flagged as "H" (High) or "L" (Low) in the Data Listings if the parameter is outside the normal range.

The ECG results will be listed per subject. Any comment on abnormal results will also be provided. Abnormalities in physical examination, ECG, clinical laboratory tests and vital signs will be classified in terms of clinical significance. Clinically significant abnormalities will be reported as adverse events (AEs).

AEs will be tabulated and summarized according to the MedDRA, version 24.1 or higher, and classified by SOC and PT.

All occurring TEAEs will be assigned to the last treatment administered. A separate listing of Serious Adverse Events (SAEs) will be presented, if applicable.

Incidence and frequency of TEAEs will be summarized descriptively by SOC and PT for each investigational product and overall.

#### 11. PRESENTATION OF RESULTS

## 11.1. Statistical Output Specification

Tables will be generated as Rich Text Files (\*.rtf) from SAS<sup>®</sup>.

Figures and Analysis Outputs will be generated as \*.docx files, exported from Phoenix WinNonlin<sup>®</sup> and/or SAS<sup>®</sup>.

In-text Tables and Figures will preferably be prepared in portrait format. Listings will preferably be prepared in landscape format.

The CSR will be written according to BlueClinical SOPs and templates for reporting bioavailability/bioequivalence trials.

## 11.2. Planned Tables, Figures, and Subject Data Listings

The planned Tables, Figures, and Individual Data Listings for the CSR are listed below.

# 11.2.1. In-text Tables and Figures

For CSR Synopsis:

The following Tables will be produced for direct insertion in the Synopsis of the CSR:

#### Title

#### PART 1

Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect)

1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect)

Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect)

1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect)

Total Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect)

Free Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect)

Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub>

1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0:t}$ 

Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$ 

#### Title

1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0\text{-t}}$ 

Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0\text{-t}}$ 

1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0-1}$ 

Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$ 

1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{04}$ 

Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub>

Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0\text{-t}}$ 

Total Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0\text{-t}}$ 

Free Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0\text{-}t}$ 

The following Figures will be produced for direct insertion in the Synopsis of the CSR:

# Legend

# PART 1

Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A –

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

| - | | | | | • |
|---|---|---|---|---|---|
| | • | a | Δ | n | |
| _ | | z | · | ш | u |

Linear Scale; B – Semi-Logarithmic Scale

1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

### For CSR Body Text:

The following Tables and Figures will be produced for direct insertion in the body text of the CSR:

| In-text Tables | Title |
|---|---|
| PART 1 | |
| Table 1.A. | Study Flow-Chart – Part 1 |
| Table 1.B. | Identity of Investigational Products – Part 1 |
| Table 1.C. | Summary of Exposure to Treatment – Part 1 |
| Table 1.D. | Summary of Subjects Disposition – Part 1 |
| Table 1.E.1. | Summary of Demographic Data of Pharmacokinetic Analysis Populations |
| Table 1.E.2. | Summary of Demographic Data of Drug-Drug Interaction Comparable<br>Bioavailability Analysis Populations – Effect of Givinostat on Midazolam IV |
| Table 1.E.3. | Summary of Demographic Data of Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Populations – Effect of Givinostat on Oral |
| | Midazolam |
| Table 1.E.4. | Summary of Demographic Data of Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Populations – Effect of Givinostat on Dabigatran |
| | Etexilate |
| Table 1.F.1. | Midazolam: Summary Statistics of the Pharmacokinetic Parameters |
| | Following Administration of Midazolam IV Alone (Day 1) and Co- |
| | Administration of Midazolam IV and Givinostat (Day 6 – Potential |
| | Inhibitory Effect, and Day 17 – Potential Inducing Effect) |
| Table 1.F.2. | 1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic |
| | Parameters Following Administration of Midazolam IV Alone (Day 1) and |
| | Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential |

| In-text Tables | Title |
|---|---|
| | Inhibitory Effect, and Day 17 – Potential Inducing Effect) |
| Table 1.G.1. | Midazolam: Summary Statistics of the Pharmacokinetic Parameters |
| | Following Administration of Oral Midazolam Alone (Day 2) and Co- |
| | Administration of Oral Midazolam and Givinostat (Day 7 – Potential |
| | Inhibitory Effect, and Day 18 – Potential Inducing Effect) |
| Table 1.G.2. | 1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic |
| | Parameters Following Administration of Oral Midazolam Alone (Day 2) and |
| | Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential |
| | Inhibitory Effect, and Day 18 – Potential Inducing Effect) |
| Table 1.H.1. | Total Dabigatran: Summary Statistics of the Pharmacokinetic Parameters |
| | Following Administration of Dabigatran Etexilate Alone (Day 1) and Co- |
| | Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential |
| | Inhibitory Effect, and Day 17 – Potential Inducing Effect) |
| Table 1.H.2. | Free Dabigatran: Summary Statistics of the Pharmacokinetic Parameters |
| | Following Administration of Dabigatran Etexilate Alone (Day 1) and Co- |
| | Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential |
| | Inhibitory Effect, and Day 17 – Potential Inducing Effect) |
| Table 1.I.1. | Midazolam: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.I.2. | 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.J.1. | Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics |
| | of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric |
| | Least Square Means, Geometric Least Square Means Ratio and |
| | Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.J.2. | 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the |
| | Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.K.1. | Midazolam: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.K.2. | 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.L.1. | Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics |
| | of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric |
| | Least Square Means, Geometric Least Square Means Ratio and |
| | Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.L.2. | 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the |
| | Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |



| In-text Tables | Title |
|---|---|
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.M.1. | Total Dabigatran: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.M.2. | Free Dabigatran: Potential Inhibitory Effect of Givinostat on the |
| | Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.N.1. | Total Dabigatran: Potential Induction Effect of Givinostat on the |
| | Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.N.2. | Free Dabigatran: Potential Induction Effect of Givinostat on the |
| | Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of |
| | Variation, Geometric Least Square Means, Geometric Least Square Means |
| | Ratio and Corresponding 90% Confidence Interval for C <sub>max</sub> and AUC <sub>0-t</sub> |
| Table 1.O.1. | Summary of Treatment-Emergent Adverse Events (TEAEs) – All TEAEs |
| Table 1.O.2. | Summary of Treatment-Emergent Adverse Events (TEAEs) – Drug-Related |
| | TEAEs |
| Table 1.O.3. | Summary of Treatment-Emergent Adverse Events (TEAEs) – |
| | Inhibition/Induction Drug-Related TEAEs |

| In-text Figures | Legend |
|---|---|
| PART 1 | |
| Figure 1.A.1. | Midazolam: Geometric Mean (95% CI) Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale |
| Figure 1.A.2. | Midazolam: Geometric Mean (95% CI) Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale |
| Figure 1.B.1. | 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration<br>Versus Time Profiles Following Administration of Midazolam IV Alone<br>(Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale |
| Figure 1.B.2. | 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration<br>Versus Time Profiles Following Administration of Midazolam IV Alone<br>(Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale |
| Figure 1.C.1. | Midazolam: Geometric Mean (95% CI) Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear Scale |
| Figure 1.C.2. | Midazolam: Geometric Mean (95% CI) Plasma Concentration Versus Time |

| In-text Figures | Legend |
|---|---|
| - teat Figures | Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co- |
| | Administration of Oral Midazolam and Givinostat (Day 7 – Potential |
| | Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi- |
| | Logarithmic Scale |
| Figure 1.D.1. | 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration |
| | Versus Time Profiles Following Administration of Oral Midazolam Alone |
| | (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – |
| | Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear |
| | Scale |
| Figure 1.D.2. | 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration |
| | Versus Time Profiles Following Administration of Oral Midazolam Alone |
| | (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – |
| | Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi- |
| | Logarithmic Scale |
| Figure 1.E.1. | Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration Versus |
| | Time Profiles Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – |
| | Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear |
| E' 1 E 0 | Scale |
| Figure 1.E.2. | Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration Versus |
| | Time Profiles Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – |
| | Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi- |
| Figure 1.F.1. | Logarithmic Scale Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration <i>Versus</i> |
| riguic 1.1.1. | Time Profiles Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – |
| | Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear |
| | Scale |
| Figure 1.F.2. | Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration Versus |
| | Time Profiles Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – |
| | Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi- |
| | Logarithmic Scale |
| Figure 3.A.4. | Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time |
| | Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day |
| | 13) – Semi-Logarithmic Scale |
| Figure 3.A.5. | Givinostat: Geometric Mean (95% CI) Trough Plasma Concentration Versus |
| | Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 |
| | to Day 13) – Linear Scale |
| Figure 3.B.1. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.B.2. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic |
| D' 0.D.0 | Scale |
| Figure 3.B.3. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma |

| In-text Figures | Legend |
|---|---|
| Ŭ | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.B.4. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.B.5. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Trough Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.C.1. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.C.2. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic |
| | Scale |
| Figure 3.C.3. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.C.4. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.C.5. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Trough Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| E. 0.D.1 | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.D.1. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| Figure 2 D 2 | Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.D.2. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma |
| | Concentration <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic |
| | Scale |
| Figure 3.D.3. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma |
| riguic 3.D.3. | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.D.4. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma |
| 1 igure 5.15.4. | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.D.5. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Trough Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.E.1. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.E.2. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Single-Dose (Day 1) and |
| | Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic |
| | Scale |
| Figure 3.E.3. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma |

| In-text Figures | Legend |
|---|---|
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.E.4. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.E.5. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Trough Plasma |
| | Concentration Versus Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.F.1. | Givinostat: Geometric Mean (95% CI) of Urinary Excretion Versus Time |
| | Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) |
| | Administration of Givinostat – Linear Scale |
| Figure 3.F.2. | Givinostat: Geometric Mean (95% CI) of Cumulative Amount Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.G.1. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.G.2. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Cumulative |
| | Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.H.1. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.H.2. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Cumulative |
| | Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.I.1. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.I.2. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Cumulative |
| | Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.J.1. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.J.2. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Cumulative |
| | Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |

# 11.2.2. Tables, Figures and Graphs Referred to But Not Included in the Text (Section 14 of CSR)

At least the following Tables and Figures should be produced for Section 14 of the CSR. If necessary, additional Tables and Figures should be prepared.

The following Tables and Figures will be compiled in a document, to be considered as Section 14 (Tables, Figures and Graph Referred To But Not Included in the Text) of the CSR.

| End of Toyt | |
|---|---|
| End-of-Text | Title |
| Tables | |
| <u>14.1. PART 1</u> | |
| 14.1.1. DEMOG | RAPHIC DATA – PART 1 |
| 14.1.1.1. | Demographic Data – Part 1 Safety Analysis Population |
| 14.1.1.2. | Demographic Data – Part 1 Pharmacokinetic Analysis Population |
| 14.1.1.3. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inhibitory Effect of Givinostat on Midazolam IV |
| 14.1.1.4. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inhibitory Effect of Givinostat on Oral Midazolam |
| 14.1.1.5. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inhibitory Effect of Givinostat on |
| | Dabigatran |
| 14.1.1.6. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inducing Effect of Givinostat on |
| | Midazolam IV |
| 14.1.1.7. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inducing Effect of Givinostat on |
| | Oral Midazolam |
| 14.1.1.8. | Demographic Data – Part 1 Drug-Drug Interaction Comparable |
| | Bioavailability Analysis Population – Inducing Effect of Givinostat on |
| | Dabigatran |
| 14.1.1.9. | Subjects Prematurely Discontinued After First Dosing |
| | ACOKINETIC DATA – PART 1 |
| 14.1.2.1. | Deviations from Blood Sampling Schedule |
| 14.1.2.1.1. | Deviations from Blood Sampling Schedule |
| 14.1.2.1.1.<br>14.1.2.1.2. | |
| | Deviations from Blood Sampling Schedule |
| 14.1.2.1.2. | Deviations from Blood Sampling Schedule Missing Blood Samples |
| 14.1.2.1.2.<br>14.1.2.1.3. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br><b>14.1.2.2.</b> | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2.<br>14.1.2.2.3. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2.<br>14.1.2.2.3. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2.<br>14.1.2.2.3. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and |
| 14.1.2.1.2.<br>14.1.2.1.3.<br>14.1.2.2.<br>14.1.2.2.1.<br>14.1.2.2.2.<br>14.1.2.2.3.<br>14.1.2.2.4.<br>14.1.2.2.5. | Deviations from Blood Sampling Schedule Missing Blood Samples Other Important Protocol Deviations Plasma Concentrations Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) |

| End-of-Text | Title |
|---|---|
| Tables | |
| 14.1.2.2.7. | Midazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Administration of Oral Midazolam Alone (Day 2) |
| 14.1.2.2.8. | Midazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Oral Midazolam and |
| | Givinostat (Day 7) |
| 14.1.2.2.9. | Midazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Oral Midazolam and |
| | Givinostat (Day 18) |
| 14.1.2.2.10. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Administration of Oral Midazolam Alone (Day 2) |
| 14.1.2.2.11. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Oral Midazolam and |
| | Givinostat (Day 7) |
| 14.1.2.2.12. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Oral Midazolam and |
| | Givinostat (Day 18) |
| 14.1.2.2.13. | Total Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) |
| 14.1.2.2.14. | Total Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Dabigatran Etexilate and |
| | Givinostat (Day 6) |
| 14.1.2.2.15. | Total Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Dabigatran Etexilate and |
| | Givinostat (Day 17) |
| 14.1.2.2.16.<br>14.1.2.2.17. | Free Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Administration of Dabigatran Etexilate Alone (Day |
| | 1) |
| | Free Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Dabigatran Etexilate and |
| | Givinostat (Day 6) |
| 14.1.2.2.18. | Free Dabigatran: Individual Data and Descriptive Statistics of Plasma |
| | Concentrations Following Co-Administration of Dabigatran Etexilate and |
| | Givinostat (Day 17) |
| 14.1.2.3. | Pharmacokinetic Parameters |
| 14.1.2.3.1. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic |
| | Parameters Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.3.2. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic |
| | Parameters Following Co-Administration of Midazolam IV and Givinostat |
| | (Day 6) |
| 14.1.2.3.3. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic |
| | Parameters Following Co-Administration of Midazolam IV and Givinostat |
| | (Day 17) |
| 14.1.2.3.4. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of |
| | Pharmacokinetic Parameters Following Administration of Midazolam IV |
| | Alone (Day 1) |
| End-of-Text<br>Tables | Title | | | |
|---|---|--|--|--|
| 14.1.2.3.5. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of<br>Pharmacokinetic Parameters Following Co-Administration of Midazolam IV<br>and Givinostat (Day 6) | | | |
| 14.1.2.3.6. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of<br>Pharmacokinetic Parameters Following Co-Administration of Midazolam IV<br>and Givinostat (Day 17) | | | |
| 14.1.2.3.7. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic<br>Parameters Following Administration of Oral Midazolam Alone (Day 2) | | | |
| 14.1.2.3.8. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 7) | | | |
| 14.1.2.3.9. | Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 18) | | | |
| 14.1.2.3.10. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of<br>Pharmacokinetic Parameters Following Administration of Oral Midazolam<br>Alone (Day 2) | | | |
| 14.1.2.3.11. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of<br>Pharmacokinetic Parameters Following Co-Administration of Oral<br>Midazolam and Givinostat (Day 7) | | | |
| 14.1.2.3.12. | 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 18) | | | |
| 14.1.2.3.13. | Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) | | | |
| 14.1.2.3.14. | Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) | | | |
| 14.1.2.3.15. | Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) | | | |
| 14.1.2.3.16. | Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) | | | |
| 14.1.2.3.17. | Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) | | | |
| 14.1.2.3.18. | Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) | | | |
| 14.1.2.3.19. | Midazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for C <sub>max</sub> | | | |
| 14.1.2.3.20. | Midazolam IV Alone (Day 1) Individual Ratios for C <sub>max</sub> Midazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to- Midazolam IV Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> | | | |
| 14.1.2.3.21. | 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for C <sub>max</sub> | | | |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.1.2.3.22. | 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day |
| 14.1.2.3.22. | 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.23. | Midazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to- |
| 14.1.2.3.23. | · · |
| 14 1 2 2 24 | Midazolam IV Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.24. | Midazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to- |
| 1410205 | Midazolam IV Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.25. | 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day |
| | 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.26. | 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day |
| | 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.27. | Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to- |
| | Oral Midazolam Alone (Day 2) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.28. | Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to- |
| | Oral Midazolam Alone (Day 2) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.29. | 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat |
| | (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.30. | 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat |
| | (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.31. | Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 18)-to- |
| | Oral Midazolam Alone (Day 2) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.32. | Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 18)-to- |
| | Oral Midazolam Alone (Day 2) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.33. | 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat |
| | (Day 18)-to-Oral Midazolam Alone (Day 2) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.34. | 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat |
| | (Day 18)-to-Oral Midazolam Alone (Day 2) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.35. | Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat ( |
| | 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.36. | Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (D |
| | 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.37. | Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.38. | Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.39. | Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.40. | Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.3.41. | Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for C <sub>max</sub> |
| 14.1.2.3.42. | Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day |
| | 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for AUC <sub>0-t</sub> |
| 14.1.2.4. | Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| 14.1.2.4.1. | Midazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation Following |
| | Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.4.2. | Midazolam: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation Following |
| | Co-Administration of Midazolam IV and Givinostat (Day 6) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.1.2.4.3. | Midazolam: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation Following |
| | Co-Administration of Midazolam IV and Givinostat (Day 17) |
| 14.1.2.4.4. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation |
| | Following Administration of Midazolam IV Alone (Day 1) |
| 14.1.2.4.5. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation |
| | Following Co-Administration of Midazolam IV and Givinostat (Day 6) |
| 14.1.2.4.6. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation Following Co-Administration of Midazolam IV and Givinostat (Day 17) |
| 14.1.2.4.7. | Midazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation Following Administration of Oral Midazolam Alone (Day 2) |
| 14.1.2.4.8. | Midazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 7) |
| 14.1.2.4.9. | Midazolam: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 18) |
| 14.1.2.4.10. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Administration of Oral Midazolam Alone (Day 2) |
| 14.1.2.4.11. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for $\lambda_z$ Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 7) |
| 14.1.2.4.12. | 1-Hydroxymidazolam: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Co-Administration of Oral Midazolam and Givinostat (Day 18) |
| 14.1.2.4.13. | Total Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Administration of Dabigatran Etexilate Alone (Day 1) |
| 14.1.2.4.14. | Total Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) |
| 14.1.2.4.15. Total Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estim | |
| | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) |
| 14.1.2.4.16. | Free Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Administration of Dabigatran Etexilate Alone (Day 1) |
| 14.1.2.4.17. | Free Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Co-Administration of Dabigatran Etexilate Co-Administered and |
| | Givinostat (Day 6) |
| 14.1.2.4.18. | Free Dabigatran: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| | Following Co-Administration of Dabigatran Etexilate Co-Administered and |
| | Givinostat (Day 17) |
| | DATA – PART 1 |
| 14.1.3.1. | Adverse Events |
| 14.1.3.1.1. | Pre-Treatment Adverse Events |
| 14.1.3.1.2. | Treatment-Emergent Adverse Events (I) |
| 14.1.3.1.3. | Treatment-Emergent Adverse Events (II) |
| 14.1.3.2. | Vital Signs |
| 14.1.3.2.1. | Descriptive Statistics of Vital Signs Parameters |
| 14.1.3.2.2. | Descriptive Statistics of Change from Baseline of Vital Signs Parameters |
| 14.1.3.2.3. | Shifts in Vital Signs Parameters |
| 14.1.3.3. | 12-Lead ECG |
| 14.1.3.3.1. | Descriptive Statistics of 12-Lead ECG Parameters |

| End-of-Text | Title |
|---|---|
| Tables | |
| 14.1.3.3.2. | Descriptive Statistics of Change from Baseline of 12-Lead ECG Parameters |
| 14.1.3.3.3. | Shifts in 12-Lead ECG Parameters |
| 14.1.3.4. | Hematology |
| 14.1.3.4.1. | Descriptive Statistics of Hematology Parameters |
| 14.1.3.4.2. | Descriptive Statistics of Change from Baseline of Hematology Parameters |
| 14.1.3.4.3. | Shifts in Hematology Parameters |
| 14.1.3.5. | Biochemistry |
| 14.1.3.5.1. | Descriptive Statistics of Biochemistry Parameters |
| 14.1.3.5.2. | Descriptive Statistics of Change from Baseline of Biochemistry Parameters |
| 14.1.3.5.3. | Shifts in Biochemistry Parameters |
| 14.1.3.6. | Coagulation |
| 14.1.3.6.1. | Descriptive Statistics of Coagulation Parameters |
| 14.1.3.6.2. | Descriptive Statistics of Change from Baseline of Coagulation Parameters |
| 14.1.3.6.3. | Shifts in Coagulation Parameters |
| 14.1.3.7. | Urinalysis |
| 14.1.3.7.1. | Descriptive Statistics of Urinalysis Parameters |
| 14.1.3.7.2. | Descriptive Statistics of Change from Baseline of Urinalysis Parameters |
| 14.1.3.7.3. | Shifts in Urinalysis Parameters |
| 14.1.3.8. | Body Weight |
| 14.1.3.8.1. | Descriptive Statistics of Body Weight |
| 14.1.3.8.2. | Descriptive Statistics of Body Weight – Male Subjects |
| 14.1.3.8.3. | Descriptive Statistics of Body Weight – Female Subjects |
| 14.1.3.8.4. | Descriptive Statistics of Change from Baseline of Body Weight |
| 14.1.3.8.5. | Descriptive Statistics of Change from Baseline of Body Weight – Male Subjects |
| 14.1.3.8.6. | Descriptive Statistics of Change from Baseline of Body Weight – Female Subjects |

| End-of-Text | Title |
|---|---|
| Figures | |
| 14.1. PART 1 | |
| 14.1.2. PHARMA | COKINETIC DATA – Part 1 |
| 14.1.2.5. | Plasma Concentration Versus Time Profiles of All Subjects |
| 14.1.2.5.1. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Administration of Midazolam IV Alone (Day 1) – Linear Scale |
| 14.1.2.5.2. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Co-Administration of Midazolam IV and Givinostat (Day 6) |
| 14.1.2.5.3. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Co-Administration of Midazolam IV and Givinostat (Day 17) |
| 14.1.2.5.4. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| | Subjects Following Administration of Midazolam IV Alone (Day 1) – Linear |
| | Scale |

| End-of-Text | Title |
|---|---|
| Figures | |
| 14.1.2.5.5. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| 11.1.2.3.3. | Subjects Following Co-Administration of Midazolam IV and Givinostat (Day |
| | 6) |
| 14.1.2.5.6. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| | Subjects Following Co-Administration of Midazolam IV and Givinostat (Day |
| | 17) |
| 14.1.2.5.7. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Administration of Oral Midazolam Alone (Day 2) – Linear Scale |
| 14.1.2.5.8. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Co-Administration of Oral Midazolam and Givinostat (Day 7) |
| 14.1.2.5.9. | Midazolam: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Co-Administration of Oral Midazolam and Givinostat (Day 18) |
| 14.1.2.5.10. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| | Subjects Following Administration of Oral Midazolam Alone (Day 2) – |
| | Linear Scale |
| 14.1.2.5.11. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| | Subjects Following Co-Administration of Oral Midazolam and Givinostat |
| | (Day 7) |
| 14.1.2.5.12. | 1-Hydroxymidazolam: Plasma Concentration Versus Time Profiles of All |
| | Subjects Following Co-Administration of Oral Midazolam and Givinostat |
| | (Day 18) |
| 14.1.2.5.13. | Total Dabigatran: Plasma Concentration Versus Time Profiles of All Subjects |
| | Following Administration of Dabigatran Etexilate Alone (Day 1) – Linear |
| | Scale |
| 14.1.2.5.14. | Total Dabigatran: Plasma Concentration Versus Time Profiles of All Subjects |
| 1410515 | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) |
| 14.1.2.5.15. | Total Dabigatran: Plasma Concentration <i>Versus</i> Time Profiles of All Subjects |
| | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day |
| 14.1.2.5.16. | 17) |
| 14.1.2.3.16. | Free Dabigatran: Plasma Concentration <i>Versus</i> Time Profiles of All Subjects Following Administration of Dabigatran Etexilate Alone (Day 1) – Linear |
| | Scale |
| 14.1.2.5.17. | Free Dabigatran: Plasma Concentration <i>Versus</i> Time Profiles of All Subjects |
| 14.1.2.3.17. | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) |
| 14.1.2.5.18. | Free Dabigatran: Plasma Concentration Versus Time Profiles of All Subjects |
| 11.1.2.3.10. | Following Co-Administration of Dabigatran Etexilate and Givinostat (Day |
| | 17) |
| 14.1.2.6. | Individual Plasma Concentration Versus Time Profiles |
| 14.1.2.6.1. | Midazolam: Individual Plasma Concentration Versus Time Profiles Following |
| | Administration of Midazolam IV Alone (Day 1) and Co-Administration of |
| | Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and I |
| | 17 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.2. | Midazolam: Individual Plasma Concentration Versus Time Profiles Following |
| | Administration of Midazolam IV Alone (Day 1) and Co-Administration of |
| | Midazolam IV and Givinostat (Day 6 - Potential Inhibitory Effect, and Day |
| | 17 – Potential Inducing Effect) – Semi-Logarithmic Scale |

| End-of-Text<br>Figures | Title |
|---|---|
| 14.1.2.6.3. | 1-Hydroxymidazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.4. | 1-Hydroxymidazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale |
| 14.1.2.6.5. | Midazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.6. | Midazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi-Logarithmic Scale |
| 14.1.2.6.7. | 1-Hydroxymidazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.8. | 1-Hydroxymidazolam: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi-Logarithmic Scale |
| 14.1.2.6.9. | Total Dabigatran: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.10. | Total Dabigatran: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co- Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi- Logarithmic Scale |
| 14.1.2.6.11. | Free Dabigatran: Individual Plasma Concentration <i>Versus</i> Time Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale |
| 14.1.2.6.12. | Free Dabigatran: Individual Plasma Concentration <i>Versus</i> Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale |

# 11.2.3. List of Subject Data Listings (Section 16.2 of CSR)

The following Data Listings will be produced for Section 16.2. Subject Data Listings of the CSR.

If necessary, additional Data Listings should be prepared.

| Listing No. | Title |
|---|---|
| 16.2. SUBJECTS | S DATA LISTING |
| 16.2.1. Part 1 | |
| 16.2.1.1. | Subject Disposition |
| 16.2.1.1.1. | Subject Disposition |
| 16.2.1.2. | Protocol Deviations |
| 16.2.1.2.1. | Blood Sampling Times Deviations |
| 16.2.1.2.2. | Other Protocol Deviations |
| 16.2.1.3. | Excluded Data from the Pharmacokinetic Analysis |
| 16.2.1.3.1. | Plasma Concentrations |
| 16.2.1.3.1.1. | Midazolam: Individual Data of Plasma Concentrations Following |
| | Administration of Midazolam IV |
| 16.2.1.3.1.2. | 1-Hydroxymidazolam: Individual Data of Plasma Concentrations Following |
| | Administration of Midazolam IV |
| 16.2.1.3.1.3. | Midazolam: Individual Data of Plasma Concentrations Following |
| | Administration of Oral Midazolam |
| 16.2.1.3.1.4. | 1-Hydroxymidazolam: Individual Data of Plasma Concentrations Following |
| | Administration of Oral Midazolam |
| 16.2.1.3.1.5. | Total Dabigatran: Individual Data of Plasma Concentrations Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.3.1.6. | Free Dabigatran: Individual Data of Plasma Concentrations Following |
| Administration of Dabigatran Etexilate | |
| 16.2.1.3.2. | Plasma Concentration Versus Time Profiles |
| 16.2.1.3.2.1. | Midazolam: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Midazolam IV – Linear Scale |
| 16.2.1.3.2.2. | Midazolam: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Midazolam IV – Semi-Logarithmic Scale |
| 16.2.1.3.2.3. | 1-Hydroxymidazolam: Individual Plasma Concentration Versus Time |
| | Profiles Following Administration of Midazolam IV – Linear Scale |
| 16.2.1.3.2.4. | 1-Hydroxymidazolam: Individual Plasma Concentration Versus Time |
| | Profiles Following Administration of Midazolam IV – Semi-Logarithmic |
| | Scale |
| 16.2.1.3.2.5. | Midazolam: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Oral Midazolam – Linear Scale |
| 16.2.1.3.2.6. | Midazolam: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Oral Midazolam – Semi-Logarithmic Scale |
| 16.2.1.3.2.7. | |
| | Profiles Following Administration of Oral Midazolam – Linear Scale |
| 16.2.1.3.2.8. | 1-Hydroxymidazolam: Individual Plasma Concentration Versus Time |
| | Profiles Following Administration of Oral Midazolam – Semi-Logarithmic |
| | Scale |
| 16.2.1.3.2.9. | Total Dabigatran: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Dabigatran Etexilate – Linear Scale |

ITF/2357/55 Version: 1.0

| Listing No. | Title |
|---|---|
| 16.2.1.3.2.10. | Total Dabigatran: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Dabigatran Etexilate – Semi-Logarithmic Scale |
| 16.2.1.3.2.11. | Free Dabigatran: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Dabigatran Etexilate – Linear Scale |
| 16.2.1.3.2.12. | Free Dabigatran: Individual Plasma Concentration Versus Time Profiles |
| | Following Administration of Dabigatran Etexilate – Semi-Logarithmic Scale |
| 16.2.1.4. | Demographic and Other Baseline Data |
| 16.2.1.4.1. | Demographic Data |
| 16.2.1.4.2. | Fertility/Contraception |
| 16.2.1.4.2.1. | Female Fertility/Contraception |
| 16.2.1.4.2.2. | Male Fertility/Contraception |
| 16.2.1.4.3. | Drugs of Abuse, Ethanol and Cotinine |
| 16.2.1.4.4. | Viral Serology at Screening |
| 16.2.1.4.5. | Previous and Concomitant Medication |
| 16.2.1.4.6. | SARS-COV-2 Test |
| 16.2.1.5. | Compliance |
| 16.2.1.5.1. | Investigational Product Administration |
| 16.2.1.6. | Individual Pharmacokinetic Data |
| 16.2.1.6.1. | Midazolam: Individual Pharmacokinetic Data Following Administration of |
| | Midazolam IV |
| 16.2.1.6.1.1. | Midazolam: Individual Drug Concentration Data Following Administration |
| | of Midazolam IV |
| 16.2.1.6.1.2. | Midazolam: Individual Pharmacokinetic Parameters Following |
| | Administration of Midazolam IV |
| 16.2.1.6.1.3. | Midazolam: Individual Pharmacokinetic Profiles Following Administration |
| | of Midazolam IV |
| 16.2.1.6.1.4. | Midazolam: Documentation of Statistical Analysis Following Administration |
| | of Midazolam IV |
| 16.2.1.6.1.4.1. | Midazolam: Non-Compartmental Analysis Output |
| 16.2.1.6.1.4.2. | Midazolam: Non-Compartmental Analysis Plots |
| 16.2.1.6.1.4.3. | Midazolam: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.1.4.4. | Midazolam: Potential Induction Effect Analysis Output |
| 16.2.1.6.2. | 1-Hydroxymidazolam: Individual Pharmacokinetic Data Following |
| | Administration of Midazolam IV |
| 16.2.1.6.2.1. | 1-Hydroxymidazolam: Individual Drug Concentration Data Following |
| | Administration Midazolam IV |
| 16.2.1.6.2.2. | 1-Hydroxymidazolam: Individual Pharmacokinetic Parameters Following |
| | Administration of Midazolam IV |
| 16.2.1.6.2.3. | 1-Hydroxymidazolam: Individual Pharmacokinetic Profiles Following |
| | Administration of Midazolam IV |
| 16.2.1.6.2.4. | 1-Hydroxymidazolam: Documentation of Statistical Analysis Following |
| | Administration of Midazolam IV |
| 16.2.1.6.2.4.1. | 1-Hydroxymidazolam: Non-Compartmental Analysis Output |
| 16.2.1.6.2.4.2. | 1-Hydroxymidazolam: Non-Compartmental Analysis Plots |
| 16.2.1.6.2.4.3. | 1-Hydroxymidazolam: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.2.4.4. | 1-Hydroxymidazolam: Potential Induction Effect Analysis Output |
| 16.2.1.6.3. | Midazolam: Individual Pharmacokinetic Data Following Administration of |

| Listing No. | Title |
|---|---|
| _ | Oral Midazolam |
| 16.2.1.6.3.1. | Midazolam: Individual Drug Concentration Data Following Administration |
| | of Oral Midazolam |
| 16.2.1.6.3.2. | Midazolam: Individual Pharmacokinetic Parameters Following |
| | Administration of Oral Midazolam |
| 16.2.1.6.3.3. | Midazolam: Individual Pharmacokinetic Profiles Following Administration |
| | of Oral Midazolam |
| 16.2.1.6.3.4. | Midazolam: Documentation of Statistical Analysis Following Administration |
| | of Oral Midazolam |
| 16.2.1.6.3.4.1. | Midazolam: Non-Compartmental Analysis Output |
| 16.2.1.6.3.4.2. | Midazolam: Non-Compartmental Analysis Plots |
| 16.2.1.6.3.4.3. | Midazolam: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.3.4.4. | Midazolam: Potential Induction Effect Analysis Output |
| 16.2.1.6.4. | 1-Hydroxymidazolam: Individual Pharmacokinetic Data Following |
| | Administration of Oral Midazolam |
| 16.2.1.6.4.1. | 1-Hydroxymidazolam: Individual Drug Concentration Data Following |
| | Administration Oral Midazolam |
| 16.2.1.6.4.2. | 1-Hydroxymidazolam: Individual Pharmacokinetic Parameters Following |
| | Administration of Oral Midazolam |
| 16.2.1.6.4.3. | 1-Hydroxymidazolam: Individual Pharmacokinetic Profiles Following |
| | Administration of Oral Midazolam |
| 16.2.1.6.4.4. | 1-Hydroxymidazolam: Documentation of Statistical Analysis Following |
| | Administration of Oral Midazolam |
| 16.2.1.6.4.4.1. | 1-Hydroxymidazolam: Non-Compartmental Analysis Output |
| 16.2.1.6.4.4.2. | 1-Hydroxymidazolam: Non-Compartmental Analysis Plots |
| 16.2.1.6.4.4.3. | 1-Hydroxymidazolam: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.4.4.4. | 1-Hydroxymidazolam: Potential Induction Effect Analysis Output |
| 16.2.1.6.5. | Total Dabigatran: Individual Pharmacokinetic Data Following Administration |
| | of Dabigatran Etexilate |
| 16.2.1.6.5.1. | Total Dabigatran: Individual Drug Concentration Data Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.5.2. | Total Dabigatran: Individual Pharmacokinetic Parameters Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.5.3. | Total Dabigatran: Individual Pharmacokinetic Profiles Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.5.4. | Total Dabigatran: Documentation of Statistical Analysis Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.5.4.1. | Total Dabigatran: Non-Compartmental Analysis Output |
| 16.2.1.6.5.4.2. | Total Dabigatran: Non-Compartmental Analysis Plots |
| 16.2.1.6.5.4.3. | Total Dabigatran: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.5.4.4. | Total Dabigatran: Potential Induction Effect Analysis Output |
| 16.2.1.6.6. | Free Dabigatran: Individual Pharmacokinetic Data Following Administration |
| | of Dabigatran Etexilate |
| 16.2.1.6.6.1. | Free Dabigatran: Individual Drug Concentration Data Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.6.2. | Free Dabigatran: Individual Pharmacokinetic Parameters Following |
| | Administration of Dabigatran Etexilate |

| Listing No. | Title |
|---|---|
| 16.2.1.6.6.3. | Free Dabigatran: Individual Pharmacokinetic Profiles Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.6.4. | Free Dabigatran: Documentation of Statistical Analysis Following |
| | Administration of Dabigatran Etexilate |
| 16.2.1.6.6.4.1. | Free Dabigatran: Non-Compartmental Analysis Output |
| 16.2.1.6.6.4.2. | Free Dabigatran: Non-Compartmental Analysis Plots |
| 16.2.1.6.6.4.3. | Free Dabigatran: Potential Inhibitory Effect Analysis Output |
| 16.2.1.6.6.4.4. | Free Dabigatran: Potential Induction Effect Analysis Output |
| 16.2.1.7. | Adverse Event Listings (Each Subject) |
| 16.2.1.7.1. | Pre-Treatment Adverse Events |
| 16.2.1.7.2. | Treatment-Emergent Adverse Events |
| 16.2.1.7.3. | Serious Adverse Events (I) |
| 16.2.1.8. | Listings of Laboratory Measurements by Subject |
| 16.2.1.8.1. | Normal Range of Laboratory Values |
| 16.2.1.8.2. | Hematology (I) |
| 16.2.1.8.3. | Hematology (II) |
| 16.2.1.8.4. | Biochemistry (I) |
| 16.2.1.8.5. | Biochemistry (II) |
| 16.2.1.8.6. | Biochemistry (III) |
| 16.2.1.8.7. | Biochemistry (IV) |
| 16.2.1.8.8. | Biochemistry (V) |
| 16.2.1.8.9. | Coagulation |
| 16.2.1.8.10. | Urinalysis |
| 16.2.1.8.11. | Urine Microscopy |
| 16.2.1.8.12. | Pregnancy Test |
| 16.2.1.8.13. | Additional (Not Planned) Laboratory Safety Tests |
| 16.2.1.9. | Vital Signs |
| 16.2.1.10. | 12-Lead ECG |

## 12. REFERENCES

- [1] ITF/2357/55 Clinical Study Protocol, Version 1.0, 29NOV2021
- [2] Food and Drug Administration (FDA), Clinical Drug Interaction Studies Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions Guidance for Industry (2020).

### 13. APPENDICES

### APPENDIX A. Planned Tables, Figures, and Subject Data Listings

## A.1. In-text Tables and Figures – For CSR Synopsis

#### A.1.1. Part 1

### SYNOPSIS TABLES (1)

Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>1</sup>

### **SYNOPSIS TABLES (2)**

1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>1</sup>

<sup>1</sup> To be generated as follows:

| Parameter (unit) | Midazolam IV Alone<br>(Day 1)<br>(n = xx) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 6)<br>(n = xx) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 17)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | XX.XX (XX.X%) | xx.xx (xx.x%) |
| $T_{\text{max}}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| $AUC_{0-t}$ ( $<$ units $A>$ ) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $AUC_{0-\infty}$ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_{z}$ (1/h) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>½</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 1 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '#For <Parameter(s)>, n=xx, for <Investigational Product> product> roduct> ro

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

## **SYNOPSIS TABLES (3)**

Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) <sup>2</sup>

### **SYNOPSIS TABLES (4)**

1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) <sup>2</sup>

<sup>2</sup> To be generated as follows:

| Parameter (unit) | Oral Midazolam Alone<br>(Day 2)<br>(n = xx) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 7)<br>(n = xx) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 18)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| $T_{max}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | XX.XX (XX.X%) | XX.XX (XX.X%) | xx.xx (xx.x%) |
| $AUC_{0-\infty}$ ( $<$ units $A>$ ) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_{z}$ (1/h) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>1/2</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for the Part 1 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > in the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > in the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > in the pharmacokinetic parameter should be followed by the pharmacokinetic parameter should be followed

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

## **SYNOPSIS TABLES (5)**

Total Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>3</sup>

### **SYNOPSIS TABLES (6)**

Free Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>3</sup>

<sup>3</sup> To be generated as follows:

| Parameter (unit) | Dabigatran Etexilate Alone<br>(Day 1)<br>(n = xx) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 6)<br>(n = xx) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 17)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $T_{max}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | XX.XX (XX.X%) | XX.XX (XX.X%) | xx.xx (xx.x%) |
| $AUC_{0-\infty}$ ( $<$ units $A>$ ) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_{z}$ (1/h) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>1/2</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for the Part 1 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > in the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > in the pharmacokinetic parameter could not be calculated for the pharmacokinetic parameter could not be calculated for the pharmacokinetic parameter could not be calculated for the pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > in the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > in the pharmacokinetic parameter should be followed by the pharmacokinetic parameter shou

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

# **SYNOPSIS TABLES (7)**

Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>4</sup>

### **SYNOPSIS TABLES (8)**

1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>4</sup>

### <sup>4</sup> To be generated as follows:

| | _ | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Midazolam IV<br>Alone (Day 1) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 6) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | xx.xx<br>xx.xx | XX.XX<br>XX.XX | xx.xx - xx.xx $xx.xx - xx.xx$ |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Midazolam of IV Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV, performed on the Potential Inhibitory Effect of Givinostat on Midazolam IV Analysis Population.

## **SYNOPSIS TABLES (9)**

Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>5</sup>

### **SYNOPSIS TABLES (10)**

1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>5</sup>

<sup>5</sup> To be generated as follows:

| | | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Midazolam IV<br>Alone (Day 1) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 17) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | xx.xx<br>xx.xx | XX.XX<br>XX.XX | XX.XX - XX.XX<br>XX.XX - XX.XX |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Midazolam of IV Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV, performed on the Potential Induction Effect of Givinostat on Midazolam IV Analysis Population.

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## **SYNOPSIS TABLES (11)**

Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$  <sup>6</sup>

### **SYNOPSIS TABLES (12)**

1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$ 

### <sup>6</sup> To be generated as follows:

| | | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Oral Midazolam<br>Alone (Day 2) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 7) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx<br>xx.xx - xx.xx |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 7) and the Geometric LSmeans of Oral Midazolam Alone (Day 2)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam, performed on the Potential Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population.

## **SYNOPSIS TABLES (13)**

Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$ 

### **SYNOPSIS TABLES (14)**

1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>7</sup>

<sup>7</sup> To be generated as follows:

| | | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Oral Midazolam<br>Alone (Day 2) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 18) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX - XX.XX<br>XX.XX - XX.XX |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 18) and the Geometric LSmeans of Oral Midazolam Alone (Day 2)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam, performed on the Potential Induction Effect of Givinostat on Oral Midazolam Analysis Population.

### **SYNOPSIS TABLES (15)**

Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\ \delta}$ 

## **SYNOPSIS TABLES (16)**

Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>8</sup>

<sup>8</sup> To be generated as follows:

| | | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Dabigatran Etexilate<br>Alone (Day 1) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 6) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx<br>xx.xx - xx.xx |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of dabigatran etexilate, performed on the Potential Inhibitory Effect of Givinostat on Dabigatran Etexilate Analysis Population.

## **SYNOPSIS TABLES (17)**

Total Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>9</sup>

### **SYNOPSIS TABLES (18)**

Free Dabigatran: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for C<sub>max</sub> and AUC<sub>0-t</sub> <sup>9</sup>

### <sup>9</sup> To be generated as follows:

| | | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Dabigatran Etexilate<br>Alone (Day 1) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 17) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | xx.xx<br>xx.xx | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx $xx.xx - xx.xx$ |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of dabigatran etexilate, performed on the Potential Induction Effect of Givinostat on Dabigatran Etexilate Analysis Population.

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## **SYNOPSIS FIGURES (19)**

Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

### **SYNOPSIS FIGURES (20)**

1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Plot the values of midazolam or its metabolite plasma concentrations (<unitsC>) on the y axis against time (h) on the x axis.

Label x axis with 'Time (h)' and y axis with 'Midazolam Concentration (<unitsC>)' or '1-Hydroxymidazolam Concentration (<unitsC>)'.

Marks on the x axis should be from time 0 to 24 h, at intervals of 4 hours, or multiples.

Plasma concentrations marks for each blood sampling scheduled timepoint should be in (i) bordered circles (in black color) without fill for Midazolam IV Alone (Day 1), (ii) solid fill circles (in dark blue color) for the Midazolam IV Co-Administered with Givinostat (Day 6) and (iii) solid fill square (in dark red color) for the Midazolam IV Co-Administered with Givinostat (Day 17).

These guidelines should be applied on every Figure produced for pharmacokinetic results of this study.

Note: These figures will present the geometric mean concentration versus time profiles calculated for the Part 1 Pharmacokinetic Analysis Population.

## **SYNOPSIS FIGURES (21)**

Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

### **SYNOPSIS FIGURES (22)**

1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Plot the values of midazolam or its metabolite plasma concentrations (<unitsC>) on the y axis against time (h) on the x axis.

Label x axis with 'Time (h)' and y axis with 'Midazolam Concentration (<unitsC>)' or '1-Hydroxymidazolam Concentration (<unitsC>)'.

Marks on the x axis should be from time 0 to 24 h, at intervals of 4 hours, or multiples.

Plasma concentrations marks for each blood sampling scheduled timepoint should be in (i) bordered circles (in black color) without fill for Oral Midazolam Alone (Day 2), (ii) solid fill circles (in dark blue color) for the Oral Midazolam Co-Administered with Givinostat (Day 7) and (iii) solid fill square (in dark red color) for the Oral Midazolam Co-Administered with Givinostat (Day 18).

These guidelines should be applied on every Figure produced for pharmacokinetic results of this study.

Note: These figures will present the geometric mean concentration versus time profiles calculated for the Part 1 Pharmacokinetic Analysis Population.

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## **SYNOPSIS FIGURES (23)**

Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

### **SYNOPSIS FIGURES (24)**

Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect). A – Linear Scale; B – Semi-Logarithmic Scale

Plot the values of total or free dabigatran plasma concentrations (<unitsC>) on the y axis against time (h) on the x axis.

Label x axis with 'Time (h)' and y axis with 'Total Dabigatran Concentration (<unitsC>)' or 'Free Dabigatran Concentration (<unitsC>)'.

Marks on the x axis should be from time 0 to 72 h, at intervals of 4 hours, or multiples.

Plasma concentrations marks for each blood sampling scheduled timepoint should be in (i) bordered circles (in black color) without fill for Dabigatran Etexilate Alone (Day 1), (ii) solid fill circles (in dark blue color) for the Dabigatran Etexilate Co-Administered with Givinostat (Day 6) and (iii) solid fill square (in dark red color) for the Dabigatran Etexilate Co-Administered with Givinostat (Day 18).

These guidelines should be applied on every Figure produced for pharmacokinetic results of this study.

Note: These figures will present the geometric mean concentration versus time profiles calculated for the Part 1 Pharmacokinetic Analysis Population.

ITF/2357/55 Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# A.2. In-text Tables and Figures – For CSR Body Text

## A.2.1. Part 1

## Table 1.A. Study Flow-Chart – Part 1

Note: To be captured from the Clinical Study Protocol (CSP) and Amendments.

## Table 1.B. Identity of Investigational Products – Part 1

Note: To be generated by the Medical Writing (MW).

# Table 1.C. Summary of Exposure to Treatment – Part 1

| Treatment | Study Day | Number of<br>Subjects |
|---|---|---|
| Midazolam (IV) 1 mg + Dabigatram 75 mg | Day 1 | XX |
| Midazolam (Oral) 2.5 mg | Day 2 | XX |
| Givinostat 50 mg b.i.d. | Days $4-5$ | XX |
| Midazolam (IV) 1 mg + Dabigatram 75 mg + Givinostat 50 mg b.i.d. | Day 6 | XX |
| Midazolam (Oral) 2.5 mg + Givinostat 50 mg b.i.d. | Day 7 | xx |
| Givinostat 50 mg b.i.d. | Days 8 – 16 | xx |
| Midazolam (IV) 1 mg + Dabigatram 75 mg + Givinostat 50 mg b.i.d. | Day 17 | xx |
| Midazolam (Oral) 2.5 mg + Givinostat 50 mg b.i.d. | Day 18 | XX |
| Givinostat 50 mg | Day 19 | XX |

Program: <SAS Program>



Table 1.D. Summary of Subjects Disposition – Part 1

| Disposition | Number of<br>Subjects |
|---|---|
| Randomized | xx |
| Discontinued after First Dosing | XX |
| Reason | |
| - <reason></reason> | XX |
| Part 1 Safety Analysis Population | XX |
| Part 1 Pharmacokinetic Analysis Population | XX |
| Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Populations | |
| Inhibitory Effect of Givinostat on Midazolam IV Analysis Population | XX |
| Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population | XX |
| Inhibitory Effect of Givinostat on Dabigatran Analysis Population | XX |
| Inducing Effect of Givinostat on Midazolam IV Analysis Population | XX |
| Inducing Effect of Givinostat on Oral Midazolam Analysis Population | XX |
| Inducing Effect of Givinostat on Dabigatran Analysis Population | XX |
| Completed Part 1 of Study | xx |

Program: <SAS Program>

Table 1.E. Table 1.E.1. Summary of Demographic Data of Pharmacokinetic Analysis Populations

| Demography | Parameter | Pharmacokinetic Analysis<br>Population |
|---|---|---|
| Age (years) | n | XX |
| | Mean | XX |
| | SD | XX.X |
| | Median | XX |
| | Minimum | XX |
| | Maximum | XX |
| Sex, n (%) | n | XX |
| | Male | xx (xx.x%) |
| | Female | xx (xx.x%) |
| Race, n (%) | n | XX |
| | <race></race> | xx (xx.x%) |
| Weight (kg) | n | XX |
| | Mean | XX.X |
| | SD | XX.XX |
| | Median | XX.X |
| | Minimum | XX.X |
| | Maximum | XX.X |
| Height (cm) | n | XX |
| | Mean | XXX |
| | SD | XX.X |
| | Median | XXX |
| | Minimum | XXX |
| | Maximum | XXX |
| Body Mass Index (kg/m²) | n | XX |
| | Mean | XX.X |
| | SD | XX.XX |
| | Median | XX.X |
| | Minimum | XX.X |
| | Maximum | XX.X |

 $n-Number\ of\ Subjects;\ SD-Standard\ Deviation$ 

Program: <SAS Program>

Table 1.E.2. Summary of Demographic Data of Drug-Drug Interaction Comparable Bioavailability Analysis Populations – Effect of Givinostat on Midazolam IV <sup>11</sup>

Table 1.E.3. Summary of Demographic Data of Drug-Drug Interaction Comparable Bioavailability Analysis Populations – Effect of Givinostat on Oral Midazolam<sup>11</sup>

Table 1.E.4. Summary of Demographic Data of Drug-Drug Interaction Comparable Bioavailability Analysis Populations – Effect of Givinostat on Dabigatran Etexilate <sup>11</sup>

<sup>11</sup> To be generated as follows:

| Demography | Parameter | Inhibitory Effect | Inducing Effect |
|---|---|---|---|
| Age (years) | n | XX | XX |
| , | Mean | XX | XX |
| | SD | XX.X | XX.X |
| | Median | XX | XX |
| | Minimum | XX | XX |
| | Maximum | XX | XX |
| Sex, n (%) | n | XX | XX |
| | Male | xx (xx.x%) | XX (XX.X%) |
| | Female | xx (xx.x%) | xx (xx.x%) |
| Race, n (%) | n | XX | XX |
| | <race></race> | xx (xx.x%) | XX (XX.X%) |
| Weight (kg) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Maximum | XX.X | XX.X |
| Height (cm) | n | XX | XX |
| | Mean | XXX | XXX |
| | SD | XX.X | XX.X |
| | Median | XXX | XXX |
| | Minimum | XXX | XXX |
| | Maximum | XXX | XXX |
| Body Mass Index (kg/m²) | n | XX | XX |
| | Mean | XX.X | XX.X |
| | SD | XX.XX | XX.XX |
| | Median | XX.X | XX.X |
| | Minimum | XX.X | XX.X |
| | Maximum | XX.X | XX.X |

n - Number of Subjects; SD - Standard Deviation

Program: <SAS Program>

#### Table 1.F.

Table 1.F.1. Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) 12

Table 1.F.2. 1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) 12

<sup>12</sup> To be generated as follows:

| Parameter (unit) | Midazolam IV Alone<br>(Day 1)<br>(n = xx) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 6)<br>(n = xx) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 17)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | XX.XX (XX.X%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $T_{max}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| $AUC_{0-t}$ ( <unitsa>)</unitsa> | XX.XX (XX.X%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $AUC_{0-\infty}$ ( $\leq$ units $A>$ ) | XX.XX (XX.X%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| %AUC <sub>extrap</sub> (%) | XX.XX (XX.X%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $\lambda_{z}$ (1/h) | XX.XX (XX.X%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $t_{\frac{1}{2}}(h)$ | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |

n – Number of Subjects

Values are geometric mean ( $G_{mean}$ ) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the  $G_{mean}$  within square brackets

T<sub>max</sub> values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 1 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '#For <Parameter(s)>, n=xx, for <Investigational Product> product> , and n=xx, for <Investigational Product> product>'.

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### Table 1.G.

Table 1.G.1. Midazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) <sup>13</sup>

Table 1.G.2. 1-Hydroxymidazolam: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) <sup>13</sup>

<sup>13</sup> To be generated as follows:

| Parameter (unit) | Oral Midazolam Alone<br>(Day 2)<br>(n = xx) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 7)<br>(n = xx) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 18)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | XX.XX (XX.X%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $T_{max}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| $AUC_{0-t}$ ( $<$ units $A>$ ) | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $AUC_{0-\infty}$ ( $<$ units $A>$ ) | XX.XX (XX.X%) | XX.XX (XX.X%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | XX.XX (XX.X%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $\lambda_{z}$ (1/h) | xx.xx (xx.x%) | XX.XX (XX.X%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $t_{\frac{1}{2}}(h)$ | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |

n – Number of Subjects

Values are geometric mean ( $G_{mean}$ ) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the  $G_{mean}$  within square brackets

T<sub>max</sub> values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for the Part I Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part I Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '#For <Parameter(s)>, n=xx, for <Investigational Product> product>'.

#### Table 1.H.

Table 1.H.1. Total Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>14</sup>

Table 1.H.2. Free Dabigatran: Summary Statistics of the Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) <sup>14</sup>

<sup>14</sup> To be generated as follows:

| Parameter (unit) | Dabigatran Etexilate Alone (Day 1) (n = xx) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 6)<br>(n = xx) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 17)<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $T_{max}(h)$ | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| $AUC_{0-t}$ ( $\leq$ units $A>$ ) | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $AUC_{0-\infty}$ ( $\leq$ units $A>$ ) | xx.xx (xx.x%) | XX.XX (XX.X%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $\lambda_{z}$ (1/h) | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $t_{\frac{1}{2}}(h)$ | xx.xx (xx.x%) | xx.xx (xx.x%) | XX.XX (XX.X%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |

n – Number of Subjects

Values are geometric mean ( $G_{mean}$ ) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the  $G_{mean}$  within square brackets

T<sub>max</sub> values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for the Part I Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part I Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '#For <Parameter(s)>, n=xx, for <Investigational Product> product>'.

#### Table 1.I.

Table 1.I.1. Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$  15

Table 1.I.2. 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}$ 

<sup>15</sup> To be generated as follows:

| | • | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Midazolam IV<br>Alone (Day 1) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 6) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx<br>xx.xx - xx.xx |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Midazolam of IV Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV, performed on the Potential Inhibitory Effect of Givinostat on Midazolam IV Analysis Population.

#### Table 1.J.

Table 1.J.1. Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\phantom{0}16}$ 

Table 1.J.2. 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Midazolam IV: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\phantom{0}16}$ 

<sup>16</sup> To be generated as follows:

| | | Geomet | ric LSmeans | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Midazolam IV<br>Alone (Day 1) | Midazolam IV<br>Co-Administered with<br>Givinostat (Day 17) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx<br>xx.xx - xx.xx |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Midazolam IV Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Midazolam of IV Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of midazolam IV, performed on the Potential Induction Effect of Givinostat on Midazolam IV Analysis Population.

#### Table 1.K.

Table 1.K.1. Midazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{17}$ 

Table 1.K.2. 1-Hydroxymidazolam: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{\text{max}}$  and  $AUC_{0-t}^{\ \ 17}$ 

### <sup>17</sup> To be generated as follows:

| | _ | Geometi | ric LSmeans | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Oral Midazolam<br>Alone (Day 2) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 7) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx<br>xx.xx - xx.xx |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 7) and the Geometric LSmeans of Oral Midazolam Alone (Day 2)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam, performed on the Potential Inhibitory Effect of Givinostat on Oral Midazolam Analysis Population.

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### Table 1.L.

Table 1.L.1. Midazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\ 18}$ 

Table 1.L.2. 1-Hydroxymidazolam: Potential Inducing Effect of Givinostat on the Pharmacokinetics of Oral Midazolam: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\ I8}$ 

#### <sup>18</sup> To be generated as follows:

| | _ | Geometric LSmeans | | | |
|---|---|---|---|---|---|
| Parameter | Total<br>ISCV% | Oral Midazolam<br>Alone (Day 2) | Oral Midazolam<br>Co-Administered with<br>Givinostat (Day 18) | GMR (%) | 90% CI |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX - XX.XX<br>XX.XX - XX.XX |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Oral Midazolam Co-Administered with Givinostat (Day 18) and the Geometric LSmeans of Oral Midazolam Alone (Day 2)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of oral midazolam, performed on the Potential Induction Effect of Givinostat on Oral Midazolam Analysis Population.
### Table 1.M.

Table 1.M.1. Total Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\ \ 19}$ 

Table 1.M.2. Free Dabigatran: Potential Inhibitory Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{19}$ 

<sup>19</sup> To be generated as follows:

| Parameter | Total<br>ISCV% | Dabigatran Etexilate<br>Alone (Day 1) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 6) | GMR (%) | 90% CI |
|---|---|---|---|---|---|
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX - XX.XX<br>XX.XX - XX.XX |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 6) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential inhibitory effect of oral givinostat on the single-dose pharmacokinetics of dabigatran etexilate, performed on the Potential Inhibitory Effect of Givinostat on Dabigatran Etexilate Analysis Population.

#### Table 1.N.

Table 1.N.1. Total Dabigatran: Potential Induction Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{2\theta}$ 

Table 1.N.2. Free Dabigatran: Potential Induction Effect of Givinostat on the Pharmacokinetics of Dabigatran Etexilate: Total Intra-Subject Coefficient of Variation, Geometric Least Square Means, Geometric Least Square Means Ratio and Corresponding 90% Confidence Interval for  $C_{max}$  and  $AUC_{0-t}^{\ 20}$ 

<sup>20</sup> To be generated as follows:

| Parameter | Total<br>ISCV% | Dabigatran Etexilate<br>Alone (Day 1) | Dabigatran Etexilate<br>Co-Administered with<br>Givinostat (Day 17) | GMR (%) | 90% CI |
|---|---|---|---|---|---|
| C <sub>max</sub><br>AUC <sub>0-t</sub> | XX.X<br>XX.X | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | xx.xx - xx.xx $xx.xx - xx.xx$ |

Geometric LSmeans values are given in <unitsC> for Cmax and <unitsA> for AUC

GMR corresponds to the ratio of the Geometric LSmeans of Dabigatran Etexilate Co-Administered with Givinostat (Day 17) and the Geometric LSmeans of Dabigatran Etexilate Alone (Day 1)

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the results of the analysis of the potential induction effect of oral givinostat on the single-dose pharmacokinetics of dabigatran etexilate, performed on the Potential Induction Effect of Givinostat on Dabigatran Etexilate Analysis Population.



Table 1.O.

Table 1.O.1. Summary of Treatment-Emergent Adverse Events (TEAEs) – All TEAEs

| | Midazolam<br>(n = xx) | Dabigatran<br>(n = xx) | Givinostat<br>(n = xx) | Total (N = xx) |
|---|---|---|---|---|
| Number of Subjects {Nr. of TEAEs}<br>(% of Subjects) | xx {xx} (xx%) | xx {xx} (xx%) | xx {xx} (xx%) | xx {xx} (xx%) |
| MedDRA System Organ Class (SOC) Preferred Term (PT) | | | | |
| <teaes soc=""> <teaes soc=""></teaes></teaes> | | | xx {xx} (xx%)<br>xx {xx} (xx%) | |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | |
| Severity<br>Mild<br>Moderate<br>Severe | xx {xx} (xx%) | xx {xx} (xx%) | xx {xx} (xx%)<br>xx {xx} (xx%)<br>xx {xx} (xx%) | xx {xx} (xx%) |

MedDRA - Medical Dictionary for Regulatory Activities

Program: <SAS Program>

| Treatment Groups | s | Substrates Alone<br>(n = xx) | | |
|---|---|---|---|---|
| Treatment Identification | Midazolam | Dabigatran | Total | Givinostat |
| Number of Subjects {Nr. of TEAEs} (% of Subjects) | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| | (xx%) | (xx%) | (xx%) | (xx%) |
| MedDRA System Organ Class (SOC) Preferred Term (PT) | | | | |
| <teaes soc=""></teaes> | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| | (xx%) | (xx%) | (xx%) | (xx%) |
| <teaes soc=""></teaes> | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| | (xx%) | (xx%) | (xx%) | (xx%) |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | |
| Severity | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| Mild | (xx%) | (xx%) | (xx%) | (xx%) |
| Moderate | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| | (xx%) | (xx%) | (xx%) | (xx%) |
| Severe | xx {xx} | xx {xx} | xx {xx} | xx {xx} |
| | (xx%) | (xx%) | (xx%) | (xx%) |

MedDRA - Medical Dictionary for Regulatory Activities

Drug-related TEAEs are those which causality was assessed as "Reasonably Possible" by the Investigator.

Program: <SAS Program>



Table 1.O.3. Summary of Treatment-Emergent Adverse Events (TEAEs) – Inhibition/Induction Drug-Related TEAEs

| Treatment Group | s | Inhibition<br>(n = x | | | | Induction<br>(n = x | | |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Identification | Midazolan | n Dabigatraı | ı Givinostat | t Total | Midazolam | Dabigatran | ı Givinosta | t Total |
| Number of<br>Subjects {Nr. of<br>TEAEs} (% of<br>Subjects) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) | xx {xx}<br>(xx%) |
| MedDRA<br>System Organ Cla<br>Preferred Term (1 | | | | | | | | |
| <teaes soc=""></teaes> | xx {xx}<br>(xx%)<br>xx {xx}<br>(xx%) | xx {xx}<br>(xx%)<br>xx {xx}<br>(xx%) | xx {xx}<br>(xx%)<br>xx {xx}<br>(xx%) | xx {xx}<br>(xx%)<br>xx<br>{xx}<br>(xx%) | | xx {xx}<br>(xx%)<br>xx {xx}<br>(xx%) | xx {xx}<br>(xx%)<br>xx {xx}<br>(xx%) | xx {xx}<br>(xx%)<br>xx<br>{xx}<br>(xx%) |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | | | | | |
| Severity<br>Mild<br>Moderate | xx {xx}<br>(xx%)<br>xx {xx} | xx {xx}<br>(xx%)<br>xx {xx} | xx {xx}<br>(xx%)<br>xx {xx} | xx {xx}<br>(xx%)<br>xx {xx} | (xx%) | xx {xx}<br>(xx%)<br>xx {xx} | xx {xx}<br>(xx%)<br>xx {xx} | xx {xx}<br>(xx%)<br>xx {xx} |
| Severe | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX} | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX}<br>(XX%) | (XX%)<br>XX {XX}<br>(XX%) |

MedDRA – Medical Dictionary for Regulatory Activities

Drug-related TEAEs are those which causality was assessed as "Reasonably Possible" by the Investigator.

Program: <SAS Program>



Figure 1.A.1. Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale

Figure 1.A.2. Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale

Figure 1.B.1. 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale

Figure 1.B.2. 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale



Figure 1.C.1. Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear Scale

Figure 1.C.2. Midazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi-Logarithmic Scale

Figure 1.D.1. 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Linear Scale

Figure 1.D.2. 1-Hydroxymidazolam: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 – Potential Inhibitory Effect, and Day 18 – Potential Inducing Effect) – Semi-Logarithmic Scale



Figure 1.E.1. Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale

Figure 1.E.2. Total Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale

Figure 1.F.1. Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale

Figure 1.F.2. Free Dabigatran: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale

Note: To be produced according to the guidelines established for the Synopsis Figure.

- A.3. Tables, Figures and Graphs Referred to But Not Included in the Text (Section 14 of CSR)
- A.3.1. Part 1
- 14.1. PART 1
- 14.1.1. DEMOGRAPHIC DATA PART 1
- 14.1.1.1. Demographic Data Part 1 Safety Analysis Population <sup>2</sup>
- 14.1.1.2. Demographic Data Part 1 Pharmacokinetic Analysis Population <sup>2</sup>
- 14.1.1.3. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inhibitory Effect of Givinostat on Midazolam IV  $^2$
- 14.1.1.4. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inhibitory Effect of Givinostat on Oral Midazolam <sup>2</sup>
- 14.1.1.5. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inhibitory Effect of Givinostat on Dabigatran <sup>2</sup>
- 14.1.1.6. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inducing Effect of Givinostat on Midazolam IV <sup>2</sup>
- 14.1.1.7. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inducing Effect of Givinostat on Oral Midazolam <sup>2</sup>
- 14.1.1.8. Demographic Data Part 1 Drug-Drug Interaction Comparable Bioavailability Analysis Population Inducing Effect of Givinostat on Dabigatran <sup>2</sup>

<sup>2</sup> To be generated as follows:

| Subject No. | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | <male <br="">Female&gt;</male> | <race></race> | XX | xxx | XX.X | XX.X |
| ≤Insert as man | y rows as deen | ned necessary> | | | | |
| | | n | XX | XX | XX | XX |
| | | Mean | XX | XXX | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.XX | XX.XX |
| | | Median | XX | XXX | XX.X | XX.X |
| | | Minimum | XX | XXX | XX.X | XX.X |
| | | Maximum | XX | xxx | XX.X | XX.X |

 $BMI-Body\ Mass\ Index;\ n-Number\ of\ Subjects;\ SD-Standard\ Deviation$ 

Program: <SAS Program>



# 14.1.1.9. Subjects Prematurely Discontinued After First Dosing

| Subject No. | Time of Discontinuation | Last Treatment<br>Administered | Reason for Discontinuation |
|---|---|---|---|
| <subject id=""></subject> | <day#></day#> | <treatment></treatment> | <reason></reason> |
| <insert as="" as<="" many="" rows="" td=""><td>deemed necessary&gt;</td><td></td><td></td></insert> | deemed necessary> | | |

Program: <SAS Program>

### 14.1.2. PHARMACOKINETIC DATA – PART 1

## 14.1.2.1. Deviations from Blood Sampling Schedule

## 14.1.2.1.1. Deviations from Blood Sampling Schedule

| Subject No. | Day of<br>Dose | Treatment | Analyte | Planned<br>Time<br>(h:min) | Deviation (h:min) |
|---|---|---|---|---|---|
| <subject></subject> | <day #=""></day> | <treatment></treatment> | <analyte></analyte> | <planned<br>blood<br/>sampling<br/>time&gt;</planned<br> | <pre><deviation (e.g.="" <="" deviation="" difficulty="" for="" reason="" time=""> with blood sampling / Subject unavailable at scheduled time)&gt;</deviation></pre> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

### 14.1.2.1.2. Missing Blood Samples

| Subject No. | Day of<br>Dose | Treatment | Analyte | Planned Time<br>(h:min) | Reason for Missing Blood Sample |
|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <treatment></treatment> | <analyte></analyte> | <planned blood="" sampling="" time=""></planned> | <reason blood="" for="" missing="" sample=""></reason> |
| <pre><insert as="" deemed="" many="" necessary="" rows=""></insert></pre> | i | | | | |

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

# 14.1.2.1.3. Other Important Protocol Deviations

| Subject No. | Day of<br>Dose | Treatment | Analyte | Category | Description |
|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <treatment></treatment> | <analyte></analyte> | <deviation category=""></deviation> | <pre><description deviation="" of=""></description></pre> |
| <pre><insert as="" deemed="" many="" necessary="" rows=""></insert></pre> | | | | | |

Program: <SAS Program>



#### 14.1.2.2. Plasma Concentrations

- 14.1.2.2.1. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) <sup>3</sup>
- 14.1.2.2.2. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.2.3. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) <sup>3</sup>
- 14.1.2.2.4. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Midazolam IV Alone (Day 1) 3
- 14.1.2.2.5. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 6)<sup>3</sup>
- 14.1.2.2.6. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Midazolam IV and Givinostat (Day 17) 3
- 14.1.2.2.7. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Oral Midazolam Alone (Day 2) 3
- 14.1.2.2.8. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Oral Midazolam and Givinostat (Day 7) 3
- 14.1.2.2.9. Midazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Oral Midazolam and Givinostat (Day 18) $^3$
- 14.1.2.2.10. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Oral Midazolam Alone (Day 2) 3
- 14.1.2.2.11. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Oral Midazolam and Givinostat (Day 7) <sup>3</sup>
- 14.1.2.2.12. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Oral Midazolam and Givinostat (Day 18) <sup>3</sup>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.1.2.2.13. Total Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Dabigatran Etexilate Alone (Day 1) 3
- 14.1.2.2.14. Total Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.2.15. Total Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17)<sup>3</sup>
- 14.1.2.2.16. Free Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Administration of Dabigatran Etexilate Alone (Day 1) <sup>3</sup>
- 14.1.2.2.17. Free Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.2.18. Free Dabigatran: Individual Data and Descriptive Statistics of Plasma Concentrations Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) <sup>3</sup>

<sup>3</sup> To be generated as follows:

| Subject No. | Duo doso | | | | | Time Pos | st-Dose (h) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject No. | Pre-dose - | x.xx | x.xx | x.xx | X.XX | x.xx | x.xx | x.xx | x.xx | x.xx | XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX |
| <subject id=""></subject> | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| <insert as="" deemed<="" many="" rows="" td=""><td>necessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | necessary> | | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| G <sub>mean</sub> ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| G <sub>mean</sub> 95% CI Lower ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| G <sub>mean</sub> 95% CI Upper ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI Lower ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI Upper ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

BLQ – Below the Limit of Quantification (LLOQ = <LLOQ> <unitsC>) of the assay (taken as missing for the calculation of log-transformed statistics and as zero for the calculation of the remaining summary statistics)

ND - Not Done

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: These tables will present the individual data and descriptive statistics of the plasma concentrations of the Part 1 Pharmacokinetic Analysis Population.



### 14.1.2.3. Pharmacokinetic Parameters

- 14.1.2.3.1. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) 3
- 14.1.2.3.2. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Midazolam IV and Givinostat (Day 6) 3
- 14.1.2.3.3. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Midazolam IV and Givinostat (Day 17) <sup>3</sup>
- 14.1.2.3.4. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Midazolam IV Alone (Day 1) <sup>3</sup>
- 14.1.2.3.5. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Midazolam IV and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.3.6. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Midazolam IV and Givinostat (Day 17) <sup>3</sup>
- 14.1.2.3.7. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2) 3
- 14.1.2.3.8. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 7)<sup>3</sup>
- 14.1.2.3.9. Midazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 18) $^3$
- 14.1.2.3.10. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Oral Midazolam Alone (Day 2)<sup>3</sup>
- 14.1.2.3.11. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 7) <sup>3</sup>
- 14.1.2.3.12. 1-Hydroxymidazolam: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Oral Midazolam and Givinostat (Day 18) <sup>3</sup>

- 14.1.2.3.13. Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) <sup>3</sup>
- 14.1.2.3.14. Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.3.15. Total Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) <sup>3</sup>
- 14.1.2.3.16. Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate Alone (Day 1) 3
- 14.1.2.3.17. Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6) <sup>3</sup>
- 14.1.2.3.18. Free Dabigatran: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17) <sup>3</sup>

<sup>4</sup> To be generated as follows:

| Subject No. | C <sub>max</sub><br>( <unitsc>)</unitsc> | T <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>( <unitsa>)</unitsa> | AUC <sub>0-∞</sub><br>( <b><unitsa></unitsa></b> ) | %AUC <sub>extrap</sub> (%) | λ <sub>z</sub><br>(1/h) | t <sub>1/2</sub> (h) |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Insert as many rows | as deemed nec | essary> | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| A <sub>mean</sub> 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |

n – Number of Subjects;  $G_{mean}$  – Geometric Mean;  $A_{mean}$  – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation;  $G_{mean}$  95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean;  $G_{mean}$  95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean;  $G_{mean}$  95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean;  $G_{mean}$  95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC – Not Calculated **Program:** <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

\_\_\_\_\_\_

Note: These tables will present the individual data and descriptive statistics of the pharmacokinetic parameters calculated for Part 1 Pharmacokinetic Analysis Population.

14.1.2.3.19. Midazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for C<sub>max</sub> <sup>5</sup>

14.1.2.3.20. Midazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for AUC<sub>0-t</sub> <sup>5</sup>

14.1.2.3.21. 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for  $C_{max}$ <sup>5</sup>

14.1.2.3.22. 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day 6)-to-Midazolam IV Alone (Day 1) Individual Ratios for  $AUC_{0t}$ <sup>5</sup>

<sup>5</sup> To be generated as follows:

| Subject No. | Midazolam IV<br>Co-Administered and<br>Givinostat (Day 6)<br>( <units>)</units> | Midazolam IV Alone<br>(Day 1)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | XX.XX | xx.xx | xx.xx |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

14.1.2.3.23. Midazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for  $C_{max}$   $^6$ 

14.1.2.3.24. Midazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for AUC $_{0\cdot t}$   $^6$ 

14.1.2.3.25. 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for  $C_{max}$ 

14.1.2.3.26. 1-Hydroxymidazolam: Midazolam IV Co-Administered and Givinostat (Day 17)-to-Midazolam IV Alone (Day 1) Individual Ratios for AUC $_{04}$   $^6$ 

<sup>6</sup> To be generated as follows:

| Subject No. | Midazolam IV<br>Co-Administered and<br>Givinostat (Day 17)<br>( <units>)</units> | Midazolam IV Alone<br>(Day 1)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | xx.xx | xx.xx | xx.xx |

<Insert as many rows as deemed necessary>

Program: <SAS Program>



14.1.2.3.27. Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for  $C_{max}$ <sup>5</sup>

14.1.2.3.28. Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for  ${\rm AUC_{0-t}}^5$ 

14.1.2.3.29. 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for  $C_{max}$ <sup>5</sup>

14.1.2.3.30. 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat (Day 7)-to-Oral Midazolam Alone (Day 2) Individual Ratios for  $AUC_{0+}^{5}$ 

<sup>5</sup> To be generated as follows:

| Subject No. | Oral Midazolam<br>Co-Administered and<br>Givinostat (Day 7)<br>( <units>)</units> | Oral Midazolam Alone<br>(Day 2)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | XX.XX | xx.xx | XX.XX |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

14.1.2.3.32. Midazolam: Oral Midazolam Co-Administered and Givinostat (Day 18)-to-Oral Midazolam Alone (Day 2) Individual Ratios for AUC<sub>0+</sub> <sup>6</sup>

14.1.2.3.34. 1-Hydroxymidazolam: Oral Midazolam Co-Administered and Givinostat (Day 18)-to-Oral Midazolam Alone (Day 2) Individual Ratios for  $AUC_{0+}$ 

<sup>6</sup> To be generated as follows:

| Subject No. | Oral Midazolam<br>Co-Administered and<br>Givinostat (Day 18)<br>( <units>)</units> | Oral Midazolam Alone<br>(Day 2)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | xx.xx |

<Insert as many rows as deemed necessary>

Program: <SAS Program>



- 14.1.2.3.35. Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $C_{max}$ <sup>5</sup>
- 14.1.2.3.36. Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for AUC<sub>0-t</sub> <sup>5</sup>
- 14.1.2.3.37. Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $C_{max}$ <sup>5</sup>
- 14.1.2.3.38. Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 6)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $AUC_{0-t}$ <sup>5</sup>

<sup>5</sup> To be generated as follows:

| Subject No. | Dabigatran Etexilate<br>Co-Administered and<br>Givinostat (Day 6)<br>( <units>)</units> | Dabigatran Etexilate Alone<br>(Day 1)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | xx.xx | XX.XX | XX.XX |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

- 14.1.2.3.39. Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $C_{max}$
- 14.1.2.3.40. Total Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $AUC_{0t}^{\ 6}$
- 14.1.2.3.41. Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $C_{max}$ <sup>6</sup>
- 14.1.2.3.42. Free Dabigatran: Dabigatran Etexilate Co-Administered and Givinostat (Day 17)-to-Dabigatran Etexilate Alone (Day 1) Individual Ratios for  $AUC_{0+}$

<sup>6</sup> To be generated as follows:

| Subject No. | Dabigatran Etexilate<br>Co-Administered and<br>Givinostat (Day 17)<br>( <units>)</units> | Dabigatran Etexilate Alone<br>(Day 1)<br>( <units>)</units> | Ratio<br>(%) |
|---|---|---|---|
| <subject id=""></subject> | xx.xx | xx.xx | xx.xx |

<Insert as many rows as deemed necessary>

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.1.2.4. Log-Linear Regression Parameters for  $\lambda_z$  Estimation
- 14.1.2.4.1. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Midazolam IV Alone (Day 1)  $^6$
- 14.1.2.4.2. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Midazolam IV and Givinostat (Day 6)  $^6$
- 14.1.2.4.3. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Midazolam IV and Givinostat (Day 17)  $^6$
- 14.1.2.4.4. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Midazolam IV Alone (Day 1)  $^6$
- 14.1.2.4.5. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Midazolam IV and Givinostat (Day 6)  $^6$
- 14.1.2.4.6. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Midazolam IV and Givinostat (Day 17)  $^6$
- 14.1.2.4.7. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Oral Midazolam Alone (Day 2)  $^6$
- 14.1.2.4.8. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 7)  $^6$
- 14.1.2.4.9. Midazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 18)  $^6$
- 14.1.2.4.10. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Oral Midazolam Alone (Day 2)  $^6$
- 14.1.2.4.11. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 7)  $^6$
- 14.1.2.4.12. 1-Hydroxymidazolam: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Oral Midazolam and Givinostat (Day 18)  $^6$
- 14.1.2.4.13. Total Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Dabigatran Etexilate Alone (Day 1)  $^6$
- 14.1.2.4.14. Total Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6)  $^6$
- 14.1.2.4.15. Total Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17)  $^6$
- 14.1.2.4.16. Free Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Administration of Dabigatran Etexilate Alone (Day 1)  $^6$



14.1.2.4.17. Free Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Dabigatran Etexilate Co-Administered and Givinostat (Day 6) <sup>6</sup>

14.1.2.4.18. Free Dabigatran: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Co-Administration of Dabigatran Etexilate Co-Administered and Givinostat (Day 17)  $^6$ 

<sup>6</sup> To be generated as follows:

| Subject No. | Lower TLIN (h) | Upper TLIN<br>(h) | No. of Time Points | RSQ |
|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX | X.XX |

<Insert as many rows as deemed necessary>

Lower TLIN – Lower Time Point Used in Regression Analysis; Upper TLIN – Upper Time Point Used in Regression Analysis; RSQ – Goodness of Fit for the Terminal Elimination Phase

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.1.2.5. Plasma Concentration Versus Time Profiles of All Subjects
- 14.1.2.5.1. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Midazolam IV Alone (Day 1) Linear Scale
- 14.1.2.5.2. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Midazolam IV and Givinostat (Day 6)
- 14.1.2.5.3. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Midazolam IV and Givinostat (Day 17)
- 14.1.2.5.4. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Midazolam IV Alone (Day 1) Linear Scale
- 14.1.2.5.5. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Midazolam IV and Givinostat (Day 6)
- 14.1.2.5.6. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Midazolam IV and Givinostat (Day 17)
- 14.1.2.5.7. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Oral Midazolam Alone (Day 2) Linear Scale
- 14.1.2.5.8. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Oral Midazolam and Givinostat (Day 7)
- 14.1.2.5.9. Midazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Oral Midazolam and Givinostat (Day 18)
- 14.1.2.5.10. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Oral Midazolam Alone (Day 2) Linear Scale
- 14.1.2.5.11. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Oral Midazolam and Givinostat (Day 7)
- 14.1.2.5.12. 1-Hydroxymidazolam: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Oral Midazolam and Givinostat (Day 18)
- 14.1.2.5.13. Total Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Dabigatran Etexilate Alone (Day 1) Linear Scale
- 14.1.2.5.14. Total Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6)
- 14.1.2.5.15. Total Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17)
- 14.1.2.5.16. Free Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Administration of Dabigatran Etexilate Alone (Day 1) Linear Scale



- 14.1.2.5.17. Free Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 6)
- 14.1.2.5.18. Free Dabigatran: Plasma Concentration *Versus* Time Profiles of All Subjects Following Co-Administration of Dabigatran Etexilate and Givinostat (Day 17)

Note: These Figures will be extracted from Phoenix® WinNonlin® 8.2 or higher.

- 14.1.2.6. Individual Plasma Concentration Versus Time Profiles
- 14.1.2.6.1. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 Potential Inhibitory Effect, and Day 17 Potential Inducing Effect) Linear Scale
- 14.1.2.6.2. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 Potential Inhibitory Effect, and Day 17 Potential Inducing Effect) Semi-Logarithmic Scale
- 14.1.2.6.3. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 Potential Inhibitory Effect, and Day 17 Potential Inducing Effect) Linear Scale
- 14.1.2.6.4. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Alone (Day 1) and Co-Administration of Midazolam IV and Givinostat (Day 6 Potential Inhibitory Effect, and Day 17 Potential Inducing Effect) Semi-Logarithmic Scale
- 14.1.2.6.5. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 Potential Inhibitory Effect, and Day 18 Potential Inducing Effect) Linear Scale
- 14.1.2.6.6. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 Potential Inhibitory Effect, and Day 18 Potential Inducing Effect) Semi-Logarithmic Scale
- 14.1.2.6.7. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 Potential Inhibitory Effect, and Day 18 Potential Inducing Effect) Linear Scale
- 14.1.2.6.8. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Alone (Day 2) and Co-Administration of Oral Midazolam and Givinostat (Day 7 Potential Inhibitory Effect, and Day 18 Potential Inducing Effect) Semi-Logarithmic Scale
- 14.1.2.6.9. Total Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 Potential Inhibitory Effect, and Day 17 Potential Inducing Effect) Linear



#### Scale

14.1.2.6.10. Total Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale

14.1.2.6.11. Free Dabigatran: Individual Plasma Concentration *Versus* Time Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Linear Scale

14.1.2.6.12. Free Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Alone (Day 1) and Co-Administration of Dabigatran Etexilate and Givinostat (Day 6 – Potential Inhibitory Effect, and Day 17 – Potential Inducing Effect) – Semi-Logarithmic Scale

Note: These figures will be extracted from Phoenix® WinNonlin® 8.2 or higher. A figure will be produced for each subject included in the pharmacokinetic analysis population.



### 14.1.3. SAFETY DATA – PART 1

## 14.1.3.1. Adverse Events

## 14.1.3.1.1. Pre-Treatment Adverse Events

| Subject No. | SOC<br>MadDDA DT | SAE? Adverse Even | | t Date and Time<br>Maxima | | Compelitor | Medication | Outcomo |
|---|---|---|---|---|---|---|---|---|
| | MedDRA PT<br>(Reported Term) | (Yes/No) | Start | End | Severity | Causality | Required? | Outcome |
| <subject id=""></subject> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <yes no=""></yes> | DDMMMYYYY<br>hh:mm> | -DDMMMYYYY-<br>hh mm> | <a href="#"><maximal< a=""> Severity of the AE&gt;</maximal<></a> | <causality ae="" of="" the=""></causality> | <yes no=""></yes> | <outcome of<br="">the AE&gt;</outcome> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event

NK – Not Known

Program: <SAS Program>



## 14.1.3.1.2. Treatment-Emergent Adverse Events (I)

| Subject No. | No. Day of Dose Treatment MedDI | | SOC<br>ModDDA DT | DRA PT SAE? Last Treatment (Ves/No) Date and Time | | Adverse Event Date and Time | |
|---|---|---|---|---|---|---|---|
| Subject No. | | | (Reported Term) | | | Start | Start |
| <subject id=""></subject> | <day #=""></day> | <treatment></treatment> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <yes no=""></yes> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

## 14.1.3.1.3. Treatment-Emergent Adverse Events (II)

| Subject No. | Day of Dose | Treatment | SOC<br>MedDRA PT<br>(Reported Term) | Maximal Severity | Causality | Medication<br>Required? | Outcome |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <treatment></treatment> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <maximal severity<br="">of the TEAE&gt;</maximal> | <causality of="" teae="" the=""></causality> | <yes no=""></yes> | <outcome of="" teae="" the=""></outcome> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event

Program: <SAS Program>

- 14.1.3.2. Vital Signs
- 14.1.3.2.1. Descriptive Statistics of Vital Signs Parameters 9
- 14.1.3.2.2. Descriptive Statistics of Change from Baseline of Vital Signs Parameters 9
- 14.1.3.2.3. Shifts in Vital Signs Parameters 10
- 14.1.3.3. 12-Lead ECG
- 14.1.3.3.1. Descriptive Statistics of 12-Lead ECG Parameters 9
- 14.1.3.3.2. Descriptive Statistics of Change from Baseline of 12-Lead ECG Parameters 9
- 14.1.3.3.3. Shifts in 12-Lead ECG Parameters 10
- 14.1.3.4. Hematology
- 14.1.3.4.1. Descriptive Statistics of Hematology Parameters 9
- 14.1.3.4.2. Descriptive Statistics of Change from Baseline of Hematology Parameters 9
- 14.1.3.4.3. Shifts in Hematology Parameters 10
- 14.1.3.5. Biochemistry
- 14.1.3.5.1. Descriptive Statistics of Biochemistry Parameters 9
- 14.1.3.5.2. Descriptive Statistics of Change from Baseline of Biochemistry Parameters 9
- 14.1.3.5.3. Shifts in Biochemistry Parameters 10
- 14.1.3.6. Coagulation
- 14.1.3.6.1. Descriptive Statistics of Coagulation Parameters 9
- 14.1.3.6.2. Descriptive Statistics of Change from Baseline of Coagulation Parameters 9
- 14.1.3.6.3. Shifts in Coagulation Parameters 10
- 14.1.3.7. Urinalysis
- 14.1.3.7.1. Descriptive Statistics of Urinalysis Parameters 9
- 14.1.3.7.2. Descriptive Statistics of Change from Baseline of Urinalysis Parameters 9

# 14.1.3.7.3. Shifts in Urinalysis Parameters 10

# <sup>9</sup> To be generated as follows:

| Parameter | Treatment | Study Day | Protocol Time | n Mean SD | SE | Median | Minimum l | Maximum |
|---|---|---|---|---|---|---|---|---|
| <parameter (unit)=""></parameter> | <treatment></treatment> | <day></day> | <protocol time=""> <protocol time=""> <protocol time=""> <protocol time=""></protocol></protocol></protocol></protocol> | xx x.xxx x.xxx | x.xxx | x.xxx | X.XXX | X.XXX |
| Insert as many ro | ws as deemed i | necessary> | | | | | | |

n – number of subjects; SD – Standard Deviation; SE – Standard Error

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

# <sup>10</sup> To be generated as follows:

| | | | Class | | |
|---|---|---|---|---|---|
| Parameter | Study Day | Protocol Time | Baseline | Post-Baseline<br>Assessment | Nr. of Subjects |
| <parameter (unit<="" td=""><td>t)&gt; <day></day></td><td><protocol time=""></protocol></td><td><low <br="">Normal/</low></td><td><low <br="">Normal/</low></td><td>XX</td></parameter> | t)> <day></day> | <protocol time=""></protocol> | <low <br="">Normal/</low> | <low <br="">Normal/</low> | XX |
| | | <protocol time=""></protocol> | High><br><low <br="">Normal/</low> | High><br><low <br="">Normal/</low> | xx |
| <insert as="" many<="" td=""><td>rows as deemed ne</td><td>cessary&gt;</td><td>High&gt;</td><td>High&gt;</td><td></td></insert> | rows as deemed ne | cessary> | High> | High> | |

Program: <SAS Program>

## 14.1.3.8. Body Weight

- 14.1.3.8.1. Descriptive Statistics of Body Weight 9
- 14.1.3.8.2. Descriptive Statistics of Body Weight Male Subjects 9
- 14.1.3.8.3. Descriptive Statistics of Body Weight Female Subjects 9
- 14.1.3.8.4. Descriptive Statistics of Change from Baseline of Body Weight 9
- 14.1.3.8.5. Descriptive Statistics of Change from Baseline of Body Weight Male Subjects 9
- 14.1.3.8.6. Descriptive Statistics of Change from Baseline of Body Weight Female Subjects 9

<sup>9</sup> To be generated as follows:

| Visit | n | Mean | SD | SE | Median | Minimum | Maximum |
|-------------|----|-------|-------|-------|--------|---------|---------|
| <day></day> | xx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx | X.XXX |

<Insert as many rows as deemed necessary>

n – number of subjects; SD – Standard Deviation; SE – Standard Error

Program: <SAS Program>



A.4. List of Subject Data Listings (Section 16.2 of CSR)

A.4.1. **Part 1** 

16.2. SUBJECTS DATA LISTINGS

16.2.1. PART 1

16.2.1.1. Subject Disposition

16.2.1.1.1. Subject Disposition

| Screening<br>No. | Date ICF Signed | Subject<br>Eligible? | Subject Given<br>an Unique<br>Subject No.? | Unique Subject No. | Inclusion Criteria<br>Not Met | Exclusion Criteria<br>Met | Other Reason for<br>Non-Eligibility | Reason for<br>Non-<br>Randomization |
|---|---|---|---|---|---|---|---|---|
| <screening number=""></screening> | <ddmmmyyyy< td=""><td>&gt;<yes no=""></yes></td><td><yes no=""></yes></td><td><unique subject<br="">No&gt;</unique></td><td><list all="" inclusion<br="">criteria that were<br/>not met&gt;</list></td><td></td><td></td><td><list for="" non-randomization="" reason=""></list></td></ddmmmyyyy<> | > <yes no=""></yes> | <yes no=""></yes> | <unique subject<br="">No&gt;</unique> | <list all="" inclusion<br="">criteria that were<br/>not met&gt;</list> | | | <list for="" non-randomization="" reason=""></list> |

<Insert as many rows as deemed necessary>

ICF – Informed Consent Form **Program:** <SAS Program>

## 16.2.1.2. Protocol Deviations

## 16.2.1.2.1. Blood Sampling Times Deviations

| Corbined No. | T4 | Compline Time or sint | Sampling Da | Davidski ve Davase | |
|---|---|---|---|---|---|
| Subject No. | Treatment | Sampling Timepoint | Scheduled/Target | Actual | —Deviation Reason |
| <subject id=""></subject> | <treatment></treatment> | <scheduled or="" time="" unscheduled=""></scheduled> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <ddmmmyyyy<br>hh mm&gt;</ddmmmyyyy<br> | <reason deviation="" for=""></reason> |
| <insert as="" many="" row<="" td=""><td>s as deemed necessary&gt;</td><td></td><td></td><td></td><td></td></insert> | s as deemed necessary> | | | | |

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

### 16.2.1.2.2. Other Protocol Deviations

| Subject No. Protocol<br>Phase | Treatment | Category | Description | Classification |
|---|---|---|---|---|
| <subject id=""><protocol<br>Phase #&gt;</protocol<br></subject> | <treatment></treatment> | <deviation<br>Category&gt;</deviation<br> | <pre><description deviation="" of="" the=""></description></pre> | <pre><important important="" not=""></important></pre> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | |

Program: <SAS Program>



16.2.1.3. Excluded Data from the Pharmacokinetic Analysis

16.2.1.3.1. Plasma Concentrations

16.2.1.3.1.1. Midazolam: Individual Data of Plasma Concentrations Following Administration of Midazolam IV 9

16.2.1.3.1.2. 1-Hydroxymidazolam: Individual Data of Plasma Concentrations Following Administration of Midazolam IV 9

16.2.1.3.1.3. Midazolam: Individual Data of Plasma Concentrations Following Administration of Oral Midazolam 9

16.2.1.3.1.4. 1-Hydroxymidazolam: Individual Data of Plasma Concentrations Following Administration of Oral Midazolam 9

16.2.1.3.1.5. Total Dabigatran: Individual Data of Plasma Concentrations Following Administration of Dabigatran Etexilate 9

16.2.1.3.1.6. Free Dabigatran: Individual Data of Plasma Concentrations Following Administration of Dabigatran Etexilate 9

<sup>9</sup> To be generated as follows:

| Subject No. Day of Dosing | | Investigational | Due dese | | | | | Time Pos | st-Dose (h) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Product | Pre-dose | | | | | | | X.XX | X.XX | | |
| <subject id=""></subject> | <day #=""></day> | <investigational<br>Product&gt;</investigational<br> | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |

<Insert as many rows as deemed necessary>

BLO – Below the Limit of Quantification (LLOO = <LLOO> <unitsC>) of the assay

ND - Not Done

Program: <SAS Program>

- 16.2.1.3.2. Plasma Concentration Versus Time Profiles
- 16.2.1.3.2.1. Midazolam: Individual Plasma Concentration Versus Time Profiles Following Administration of Midazolam IV Linear Scale
- 16.2.1.3.2.2. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Semi-Logarithmic Scale
- 16.2.1.3.2.3. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Linear Scale
- 16.2.1.3.2.4. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Midazolam IV Semi-Logarithmic Scale
- 16.2.1.3.2.5. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Linear Scale
- 16.2.1.3.2.6. Midazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Semi-Logarithmic Scale
- 16.2.1.3.2.7. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Linear Scale
- 16.2.1.3.2.8. 1-Hydroxymidazolam: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Oral Midazolam Semi-Logarithmic Scale
- 16.2.1.3.2.9. Total Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Linear Scale
- 16.2.1.3.2.10. Total Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Semi-Logarithmic Scale
- 16.2.1.3.2.11. Free Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Linear Scale
- 16.2.1.3.2.12. Free Dabigatran: Individual Plasma Concentration *Versus* Time Profiles Following Administration of Dabigatran Etexilate Semi-Logarithmic Scale



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

Note: These Figures will be extracted from Phoenix® WinNonlin® 8.2 or higher. A figure will be produced for each subject with data excluded from the pharmacokinetic analysis.



# 16.2.1.4. Demographic and Other Baseline Data

## 16.2.1.4.1. Demographic Data

| Subject No. | Date ICF Signed | Date of Birth | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy></ddmmmyyyy> | · <mmmyyyy></mmmyyyy> | <m f=""></m> | <race></race> | xx | xxx | XX.X | XX.X |

<Insert as many rows as deemed necessary>

ICF – Informed Consent Form; BMI – Body Mass Index; M – Male; F – Female

Program: <SAS Program>



# 16.2.1.4.2. Fertility/Contraception

## 16.2.1.4.2.1. Female Fertility/Contraception

| Subject No. | Childbearing Potential? | If Yes, Birth Control Method | d Breast Feeding? | Comments |
|---|---|---|---|---|
| <subject id=""></subject> | <yes no=""></yes> | <birth control="" method=""></birth> | <yes no=""></yes> | <comments></comments> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | |

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

## 16.2.1.4.2.2. Male Fertility/Contraception

| Subject No. | Sexually Active? Agrees to Use Condom? his | | Female partner agrees to use a highly effective method of contraception? | Agree not to donate sperm<br>from first dose administration<br>until at least 90 days after the<br>last study drug administration | Comments |
|---|---|---|---|---|---|
| <subject id=""></subject> | <yes no=""></yes> | <yes no=""></yes> | <yes no=""></yes> | <yes no=""></yes> | <comments></comments> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | | |

Program: <SAS Program>


Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.4.3. Drugs of Abuse, Ethanol and Cotinine

| Subject No. | Investigation<br>Product | nal<br>Date and Tin | ne Amphetamii | nesBenzodiazepi | inesCocaine | Cannabinoids Opiates | | Ethanol | Cotinine |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <investigation< th=""><th>onal<ddmmmy< th=""><th>YYY<positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive></th></positive></th></positive></th></positive></th></ddmmmy<></th></investigation<> | onal <ddmmmy< th=""><th>YYY<positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive></th></positive></th></positive></th></positive></th></ddmmmy<> | YYY <positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive></th></positive></th></positive></th></positive> | <positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive></th></positive></th></positive> | <positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive></th></positive> | <positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive></th></positive> | <positive <="" th=""><th><positive <="" th=""><th><positive <="" th=""></positive></th></positive></th></positive> | <positive <="" th=""><th><positive <="" th=""></positive></th></positive> | <positive <="" th=""></positive> |
| - | Product> | hh:mm> | Negative> | Negative> | Negative> | Negative> | Negative> | Negative> | Negative> |

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.4.4. Viral Serology at Screening

| Subject No. | Actual Date and Time | Protocol Phase | HIV-1 & HIV-2 | Hepatitis B | Hepatitis C |
|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <qualitative value=""></qualitative> | <qualitative value=""></qualitative> | <qualitative value=""></qualitative> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | | |

HIV – Human Immunodeficiency Virus

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 16.2.1.4.5. Previous and Concomitant Medication

| Subject No. | Tuestment | Drug Name Indication | Pharmaceutical Dose (units) Frequency | Donto | Date and Time | |
|---|---|---|---|---|---|---|
| | Treatment | Drug Name<br>[ATC Code] Indication | Form Dose (units) Frequency | Route | Start | End |
| <subject id=""></subject> | <treatment></treatment> | <pre><generic <="" [xxxxxxx]="" name="" therapeutic=""> indication &gt;</generic></pre> | <pharmaceutical<dose (units)=""><frequency> Form&gt;</frequency></pharmaceutical<dose> | <route></route> | <ddmmmyyyy></ddmmmyyyy> | CDDMMMYYYY<br>or Ongoing> |

<Insert as many rows as deemed necessary>

ATC – Anatomical Therapeutic Chemical

NK - Not Known

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 16.2.1.4.6. SARS-COV-2 Test

| Subject No. | Actual Date | Protocol Phase | Result | If Unscheduled, Reason |
|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy></ddmmmyyyy> | <protocol phase=""></protocol> | <not detectable,="" inconclusive=""></not> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

16.2.1.5. Compliance

## 16.2.1.5.1. Investigational Product Administration

| Subject No. | Date | Actual<br>Clock Time | Investigational D<br>Product | Oose (units) | Investigational<br>Product<br>Formulation | Route of<br>Administration | Hands and<br>1Mouth Check | 150 mL of<br>? water taken? | Comments |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy<br>YY/ N/A&gt;</ddmmmyy<br> | <hh:mm a="" n=""></hh:mm> | <investigational<<br>Product&gt;</investigational<<br> | Dose (units)> | <formulation></formulation> | <route></route> | <yes a<="" n="" no="" td=""><td>&gt;<yes a="" n="" no=""></yes></td><td><comments></comments></td></yes> | > <yes a="" n="" no=""></yes> | <comments></comments> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | | | | | | |

N/A – Not Applicable

Program: <SAS Program>

#### 16.2.1.6. Individual Pharmacokinetic Data

16.2.1.6.1. Midazolam: Individual Pharmacokinetic Data Following Administration of Midazolam IV

16.2.1.6.1.1. Midazolam: Individual Drug Concentration Data Following Administration of Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.1. to 14.1.2.2.3.'

# 16.2.1.6.1.2. Midazolam: Individual Pharmacokinetic Parameters Following Administration of Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.1. to 14.1.2.3.3.'

## 16.2.1.6.1.3. Midazolam: Individual Pharmacokinetic Profiles Following Administration of Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.1. to 14.1.2.6.2.'

## 16.2.1.6.1.4. Midazolam: Documentation of Statistical Analysis Following Administration of Midazolam IV

16.2.1.6.1.4.1. Midazolam: Non-Compartmental Analysis Output

16.2.1.6.1.4.2. Midazolam: Non-Compartmental Analysis Plots

16.2.1.6.1.4.3. Midazolam: Potential Inhibitory Effect Analysis Output

16.2.1.6.1.4.4. Midazolam: Potential Induction Effect Analysis Output

# 16.2.1.6.2. 1-Hydroxymidazolam: Individual Pharmacokinetic Data Following Administration of Midazolam IV

## 16.2.1.6.2.1. 1-Hydroxymidazolam: Individual Drug Concentration Data Following Administration Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.4. to 14.1.2.2.6.'

# 16.2.1.6.2.2. 1-Hydroxymidazolam: Individual Pharmacokinetic Parameters Following Administration of Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.4. to 14.1.2.3.6.'

# 16.2.1.6.2.3. 1-Hydroxymidazolam: Individual Pharmacokinetic Profiles Following Administration of Midazolam IV

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.3. to 14.1.2.6.4.'

## 16.2.1.6.2.4. 1-Hydroxymidazolam: Documentation of Statistical Analysis Following Administration of Midazolam IV

16.2.1.6.2.4.1. 1-Hydroxymidazolam: Non-Compartmental Analysis Output

16.2.1.6.2.4.2. 1-Hydroxymidazolam: Non-Compartmental Analysis Plots

16.2.1.6.2.4.3. 1-Hydroxymidazolam: Potential Inhibitory Effect Analysis Output

16.2.1.6.2.4.4. 1-Hydroxymidazolam: Potential Induction Effect Analysis Output

#### 16.2.1.6.3. Midazolam: Individual Pharmacokinetic Data Following Administration of Oral Midazolam

## 16.2.1.6.3.1. Midazolam: Individual Drug Concentration Data Following Administration of Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.7. to 14.1.2.2.9.'

## 16.2.1.6.3.2. Midazolam: Individual Pharmacokinetic Parameters Following Administration of Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.7. to 14.1.2.3.9.'

# 16.2.1.6.3.3. Midazolam: Individual Pharmacokinetic Profiles Following Administration of Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.5. to 14.1.2.6.6.'

## 16.2.1.6.3.4. Midazolam: Documentation of Statistical Analysis Following Administration of Oral Midazolam

16.2.1.6.3.4.1. Midazolam: Non-Compartmental Analysis Output

16.2.1.6.3.4.2. Midazolam: Non-Compartmental Analysis Plots

16.2.1.6.3.4.3. Midazolam: Potential Inhibitory Effect Analysis Output

16.2.1.6.3.4.4. Midazolam: Potential Induction Effect Analysis Output

# 16.2.1.6.4. 1-Hydroxymidazolam: Individual Pharmacokinetic Data Following Administration of Oral Midazolam

## 16.2.1.6.4.1. 1-Hydroxymidazolam: Individual Drug Concentration Data Following Administration Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.10. to 14.1.2.2.12.'

# 16.2.1.6.4.2. 1-Hydroxymidazolam: Individual Pharmacokinetic Parameters Following Administration of Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.10. to 14.1.2.3.12.'

# 16.2.1.6.4.3. 1-Hydroxymidazolam: Individual Pharmacokinetic Profiles Following Administration of Oral Midazolam

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.7. to 14.1.2.6.8.'

## 16.2.1.6.4.4. 1-Hydroxymidazolam: Documentation of Statistical Analysis Following Administration of Oral Midazolam

16.2.1.6.4.4.1. 1-Hydroxymidazolam: Non-Compartmental Analysis Output

16.2.1.6.4.4.2. 1-Hydroxymidazolam: Non-Compartmental Analysis Plots

16.2.1.6.4.4.3. 1-Hydroxymidazolam: Potential Inhibitory Effect Analysis Output

16.2.1.6.4.4.4. 1-Hydroxymidazolam: Potential Induction Effect Analysis Output

# 16.2.1.6.5. Total Dabigatran: Individual Pharmacokinetic Data Following Administration of Dabigatran Etexilate

# 16.2.1.6.5.1. Total Dabigatran: Individual Drug Concentration Data Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.13. to 14.1.2.2.15.'

# 16.2.1.6.5.2. Total Dabigatran: Individual Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.13. to 14.1.2.3.15.'

# 16.2.1.6.5.3. Total Dabigatran: Individual Pharmacokinetic Profiles Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.9. to 14.1.2.6.10.'

# 16.2.1.6.5.4. Total Dabigatran: Documentation of Statistical Analysis Following Administration of Dabigatran Etexilate

16.2.1.6.5.4.1. Total Dabigatran: Non-Compartmental Analysis Output

16.2.1.6.5.4.2. Total Dabigatran: Non-Compartmental Analysis Plots

16.2.1.6.5.4.3. Total Dabigatran: Potential Inhibitory Effect Analysis Output

16.2.1.6.5.4.4. Total Dabigatran: Potential Induction Effect Analysis Output

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.6.6. Free Dabigatran: Individual Pharmacokinetic Data Following Administration of Dabigatran Etexilate

# 16.2.1.6.6.1. Free Dabigatran: Individual Drug Concentration Data Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.2.16. to 14.1.2.2.18.'

# 16.2.1.6.6.2. Free Dabigatran: Individual Pharmacokinetic Parameters Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.3.16. to 14.1.2.3.18.'

# 16.2.1.6.6.3. Free Dabigatran: Individual Pharmacokinetic Profiles Following Administration of Dabigatran Etexilate

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.1.2.6.11. to 14.1.2.6.12.'

# 16.2.1.6.6.4. Free Dabigatran: Documentation of Statistical Analysis Following Administration of Dabigatran Etexilate

16.2.1.6.6.4.1. Free Dabigatran: Non-Compartmental Analysis Output

16.2.1.6.6.4.2. Free Dabigatran: Non-Compartmental Analysis Plots

16.2.1.6.6.4.3. Free Dabigatran: Potential Inhibitory Effect Analysis Output

16.2.1.6.6.4.4. Free Dabigatran: Potential Induction Effect Analysis Output



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.7. Adverse Event Listings (Each Subject)

### 16.2.1.7.1. Pre-Treatment Adverse Events 7

### 16.2.1.7.2. Treatment-Emergent Adverse Events 7

<sup>7</sup> To be generated as follows:

| Subject No. | Day of<br>Dose | Treatment | Reported<br>Term | Serious? | Maximal<br>Severity | Causality | Action<br>Taken | Medication<br>Required? | Outcome | Adverse<br>Event Start<br>Date and<br>Time | Adverse<br>Event End<br>Date and<br>Time | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <investigational product=""></investigational> | <ae<br>Reported<br/>Term&gt;</ae<br> | <yes no=""></yes> | Moderate or<br>Severe > | Possible or<br>Reasonably<br>Possible> | Dose Not | | <fatal, not<br="">Recovered /<br/>Not<br/>Resolved,<br/>Recovered /<br/>Resolved<br/>with<br/>Sequelae,<br/>Recovering<br/>/ Resolving<br/>or<br/>Unknown&gt;</fatal,> | YYYY<br>hh:mm> | <pre><ddmmm hh="" mm="" ongoing="" or="" yyyy=""></ddmmm></pre> | <comments></comments> |

<Insert as many rows as deemed necessary>

NK - Not Known

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: The "Investigational Product" column will only be generated for Table 16.2.1.7.2. If an Adverse Event is related to Medical History, that information will be reported in 'Comments'. The "Comments" column will only be generated if there are reported comments for the adverse events.



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.7.3. Serious Adverse Events (I)

| Subject No. | Treatment | Reported Term | Reason for Seriousness | Details |
|---|---|---|---|---|
| <subject id=""></subject> | <treatment></treatment> | <ae reported="" term=""></ae> | <reason></reason> | <sae details=""></sae> |
| <insert as="" de<="" many="" rows="" td=""><td>emed necessary&gt;</td><td></td><td></td><td></td></insert> | emed necessary> | | | |

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8. Listings of Laboratory Measurements by Subject

## 16.2.1.8.1. Normal Range of Laboratory Values

| | | | | | Norm | al Range | | _ |
|---|---|---|---|---|---|---|---|---|
| | | | | Fe | male | N | <b>I</b> ale | |
| Category | Analyte | Age | Units | LLN | ULN | LLN | ULN | Qualitative |
| <category></category> | <laboratory analyte=""></laboratory> | <age interval=""></age> | <units></units> | | | | | <qualitative<br>Values&gt;</qualitative<br> |

<Insert as many rows as deemed necessary>

LLN – Lower Limit Normal; ULN – Upper Limit Normal

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.8.2. Hematology (I)

| Subject No. Actual Date Protocol and Time Phase | Hemoglob<br>(g/dL) | in RBC<br>(10^12/L) | Hematocri<br>(%) | t MCV<br>(fL) | MCH<br>(pg) | MCHC<br>(g/dL) | RDW-CV<br>(%) | Total<br>WBC<br>(10^9/L) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <pre> <subject id=""><ddmmmy<protocol< td=""><td>XX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td><td>xx</td><td>xx</td><td>XX</td><td><reason></reason></td></ddmmmy<protocol<></subject></pre> | XX | xx | XX | XX | XX | xx | xx | XX | <reason></reason> |

#### <Insert as many rows as deemed necessary>

RBC – Red Blood Cell; MCV – Mean Corpuscular Volume; MCH – Mean Corpuscular Hemoglobin; MCHC – Mean Corpuscular Hemoglobin Concentration; RDW-CV – Coefficient Variation of the Red Cell Distribution Width; WBC – White Blood Cell

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.3. Hematology (II)

| Subject No. | Actual Date<br>and Time | Protocol<br>Phase | Neutrophils<br>(10^9/L) | Eosinophils<br>(10^9/L) | Basophils<br>(10^9/L) | Lymphocyte<br>(10^9/L) | es Monocytes<br>(10^9/L) | Platelets<br>(10^9/L) | Mean Platele<br>Volume<br>(fL) | etIf<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | ODMMMY YYY hh:mm | | XX | XX | XX | XX | XX | XX | XX | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.4. Biochemistry (I)

| Subject No. | Actual Date and Time | Protocol Phase | AST<br>(IU/L) | ALT<br>(IU/L) | GGT<br>(IU/L) | LDH<br>(IU/L) | ALP<br>(IU/L) | CK<br>(IU/L) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy< td=""><td><protocol phase=""></protocol></td><td>xx</td><td>xxx</td><td>xx</td><td>xx</td><td>xx</td><td>xx</td><td><reason></reason></td></ddmmmyy<> | <protocol phase=""></protocol> | xx | xxx | xx | xx | xx | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.5. Biochemistry (II)

| Subject No. | Actual Date and Time | Protocol Phase | Creatinine<br>(mg/dL) | eGFR | Urea<br>(mg/dL) | Sodium<br>(mmol/L) | Potassium<br>(mmol/L) | Calcium<br>(mg/dL) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | <protocol phase=""></protocol> | xx | xxx | xx | xx | XX | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.6. Biochemistry (III)

| Subject No. | Actual Date<br>and Time | Protocol Phase | Magnesium<br>(mg/dL) | Glucose<br>(mg/dL) | Total<br>Cholesterol<br>(mg/dL) | Triglycerides (mg/dL) | Albumin<br>(g/dL) | Total Protein<br>(g/dL) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy<br>YY hh mm&gt;</ddmmmyy<br> | <protocol<br>Phase&gt;</protocol<br> | xx | xxx | xx | XX | xx | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.7. Biochemistry (IV)

| Subject No. | Actual Date<br>and Time | Protocol Phase | Uric Acid<br>(mg/dL) | Total Bilirubin<br>(mg/dL) | Direct<br>Bilirubin<br>(mg/dL) | Indirect<br>Bilirubin<br>(mg/dL) | TSH<br>(mIU/L) | Chloride<br>(mmol/L) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | <protocol<br>Phase&gt;</protocol<br> | xx | xxx | xx | xx | xx | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.8.8. Biochemistry (V)

| Subject No. | Actual Date<br>and Time | Protocol Phase | Amylase<br>(g/dL) | LDL<br>Cholesterol<br>(mg/dL) | HDL<br>Cholesterol<br>(mg/dL) | FSH<br>(mg/dL) | C-Reactive<br>Protein | Cystain C | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | <protocol<br>Phase&gt;</protocol<br> | XX | xxx | xx | xx | xx | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.8.9. Coagulation

| Subject No. | Actual Date and<br>Time | Protocol Phase | Prothrombin Rate<br>(%) | e Prothrombin Tim<br>(sec) | <sup>ie</sup> INR | aPTT<br>(sec) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | xx | XX.X | x.xx | XX.X | <reason></reason> |

<Insert as many rows as deemed necessary>

INR - International Normalized Ratio; aPTT - Activated Partial Thromboplastin Time

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.8.10. Urinalysis

| Subject<br>No. | Actual<br>Date and<br>Time | Protocol<br>Phase pH | Specific<br>Gravity | Protein | Hemoglobin | Glucose | Ketones | Bilirubin | Nitrites | Urobilinogen | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmm<br>MYYYY<br/>hh:mm&gt;</ddmm<br> | <protoco<br>1 Phase&gt; XX.X</protoco<br> | x.xxx | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; NCR - Not Clinically Relevant; CR - Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.11. Urine Microscopy

| Subject No. | Actual Date and<br>Time | Protocol Phase | Squamous<br>Epithelial Cells<br>(/uL) | Erythrocytes<br>(/uL) | Leukocytes<br>(/uL) | Observations | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <pre><protocol phase=""></protocol></pre> | <qualitative<br>Value&gt;</qualitative<br> | xx | xx | <observations></observations> | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.12. Pregnancy Test

| Subject No. | Actual Date and Time | Protocol Phase | Matrix | Result | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <serum or="" urine=""></serum> | <positive negative="" or=""></positive> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.13. Additional (Not Planned) Laboratory Safety Tests

| Subject No. | Actual Date and<br>Time | Protocol Phase | Investigational<br>Product | Parameter | Results | Reason |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <investigational<br>Product&gt;</investigational<br> | <parameter></parameter> | <results></results> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.9. Vital Signs

| Subject No. | Scheduled<br>Time | Actual Date<br>and Time | Protocol<br>Phase | Treatment | SBP<br>(mmHg) | DBP<br>(mmHg) | Pulse Rate<br>(beats/min) | Body<br>Temperature<br>(°C) | Respiratory<br>Rate<br>(beats/min) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <scheduled or="" time="" unscheduled=""></scheduled> | YYY hh:mm> | | <treatment></treatment> | XX | XX | XX | XX | XX | <reason></reason> |

<Insert as many rows as deemed necessary>

SBP - Systolic Blood Pressure; DBP - Diastolic Blood Pressure

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 16.2.1.10. 12-Lead ECG

| Subject No. | Scheduled<br>Time | Actual Date<br>and Time | Protocol Phase | Treatment | QTcF<br>(msec) | Result | If Abnormal,<br>Reason | If Abnormal,<br>Clinically<br>Significant? | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <scheduled<br>Time or<br/>Unscheduled&gt;</scheduled<br> | <ddmmmyy<br>YY hh:mm&gt;</ddmmmyy<br> | <protocol<br>Phase&gt;</protocol<br> | <treatment></treatment> | XXX | <abnormal <br="">Normal&gt;</abnormal> | <reason for<br="">being<br/>considered<br/>abnormal&gt;</reason> | <yes no=""></yes> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 14. ANNEXES

Annex 1: Data Blind Review Process Minute - Part 1

Annex 2: List of Subjects Dosed - Part 1